# Demande de participation à un projet de recherche médical :

**APPROUVÉ**Par CCER , 12:36, 18/07/2022

# @neurIST: informatique biomédicale intégrée pour la gestion des anévrismes cérébraux

Madame, Monsieur

Nous vous proposons de participer à notre projet de recherche.

Votre participation est entièrement libre. Toutes les données collectées dans le cadre de ce projet sont soumises à des règles strictes en matière de protection des données.

Le projet de recherche est mené par les Hôpitaux Universitaire de Genève. Nous vous en communiquerons les résultats si vous le souhaitez.

Lors d'un entretien, nous vous présenterons les éléments essentiels et répondrons à vos questions. Pour vous proposer d'ores et déjà un aperçu du projet, voici les points clés à retenir. Vous trouverez à la suite des informations complémentaires plus détaillées.

# Pourquoi menons-nous ce projet de recherche?

- Notre projet porte sur les anévrismes cérébraux qui sont des anomalies observées sur les vaisseaux sanguins irriguant notre cerveau. Les anévrismes cérébraux sont diagnostiqués par radiographie, scanners, angiographie ou IRM. L'évolution d'un anévrisme peut mener à une hémorragie potentiellement fatale ou occasionner des lésions cérébrales affectant la qualité de vie à long terme.
- Notre projet de recherche vise à déterminer les causes et les évolutions des anévrismes cérébraux afin d'améliorer leur prise en charge.
- La participation à ce projet est ouverte aux :
  - Patient·e·s chez qui un anévrisme cérébral a été diagnostiqué ;
  - Membres d'une famille chez qui des personnes liées par le sang sont affectées par un anévrisme cérébral;
  - o Personnes ne souffrant pas d'anévrisme cérébral (Volontaire sain⋅e).

# Que dois-je faire si j'accepte de participer? – Que se passe-t-il pour moi en cas de participation?

- Forme de la participation :
  - Si vous acceptez de participer à notre projet en tant que patient e diagnostiqué e avec un anévrisme cérébral, nous récolterons des informations générales vous concernant et nous vous prélèverons du sang, de la salive et des selles. Si votre anévrisme cérébral est traité, nous conserverons pour la recherche les tissus et le liquide enlevés dans le cadre de votre traitement.
  - Si vous acceptez de participer à notre projet en tant que membre d'une famille affectée par les anévrismes cérébraux ou en tant que volontaire sain·e, nous




récolterons des informations générales vous concernant et nous vous prélèverons du sang, de la salive et des selles.

- Déroulement pour les participant·e·s :
  - Si vous participez au projet en tant que patient·e: la participation à cette étude implique, en plus de votre suivi habituel, une ou plusieurs prise·s de sang, le prélèvement de salive et de selles, et un questionnaire sur votre qualité de vie que vous devrez remplir lors de visites de routine. Des informations vous concernant et concernant votre anévrisme seront relevées à partir de votre dossier hospitalier. Vous pourrez aussi être contacté·e pour fournir des informations complémentaires ou pour donner votre autorisation pour d'autres études cliniques.
  - Si vous participez au projet en tant que membre de la famille ou volontaire sain·e: la participation à cette étude implique une visite à l'hôpital pour répondre à des questions sur votre état de santé et sur votre qualité de vie, et pour effectuer une prise de sang et pour collecter de la salive et des selles. Il vous sera demandé de remplir le questionnaire sur votre qualité de vie environ tous les 5 ans. Vous pourrez aussi être contacté·e pour fournir des informations complémentaires ou pour donner votre autorisation pour d'autres études cliniques.

# Quels sont les bénéfices et les risques liés à la participation au projet ?

#### Bénéfices

- Votre participation à ce projet de recherche ne vous apportera aucun bénéfice direct.
- Par votre participation, vous contribuez à aider les futur es patient es.

# Risques et contraintes

 Les risques associés à cette étude sont ceux liés à la réalisation d'une prise de sang (risque infectieux faible, hématome) et à l'utilisation d'un réseau informatique pour le transfert des données dont la sécurité ne peut jamais être totalement garantie.

En apposant votre signature à la fin du document, vous certifiez en avoir compris le contenu et consentir librement à prendre part au projet.




#### Information détaillée

# 1. Objectif du projet et sélection des participant·e·s

Dans cette feuille d'information, notre projet de recherche est aussi simplement désigné par le terme *projet*. Si vous acceptez d'y prendre part, vous êtes *un participant/une participante au projet*.

Ce projet permettra de mieux comprendre les causes et les évolutions des anévrismes cérébraux afin d'améliorer leur prise en charge. Ce projet conduira en effet à la création d'un système informatisé d'aide à la décision pour le traitement des anévrismes cérébraux.

Nous vous sollicitons car la participation est ouverte aux :

- o Patient·e·s chez qui un anévrisme cérébral a été diagnostiqué ;
- Membres d'une famille chez qui deux personnes liées par le sang sont affectées par un anévrisme cérébral;
- Aux personnes non diagnostiquées préalablement avec un anévrisme cérébral et dont deux membres de la famille n'ont pas non plus été diagnostiqués préalablement avec un anévrisme cérébral, autrement dit toute personne ignorant avoir elle-même un antécédent d'anévrisme cérébral ou qu'un membre de sa famille lié par le sang ai un antécédent d'anévrisme cérébral : Volontaire sain·e

# 2. Informations générales sur le projet

Ce projet international regroupant plusieurs centres hospitaliers a débuté en 2006. Les études menées sur les anévrismes cérébraux suggèrent que plusieurs facteurs sont impliqués dans l'apparition et l'évolution de cette maladie. Parmi ces facteurs, nos gènes, nos protéines et notre microbiote (bactéries vivant dans notre bouche et notre système digestif) semblent jouer un rôle important. Bien qu'il ait été montré que des modifications du microbiote par l'alimentation ou la consommation d'antibiotiques influence l'évolution de diverses maladies, son rôle dans l'apparition et l'évolution des anévrismes cérébraux n'est pas clairement défini.

Pour tous les participant·e·s, nous récolterons des informations générales vous concernant et nous vous prélèverons du sang, de la salive et des selles.

Si vous participez à ce projet en tant que patient·e·s, nous récolterons également des informations concernant votre anévrisme. Lors de l'intervention pour le traitement de votre anévrisme, une partie de celui-ci pourra être prélevé, ainsi que du liquide céphalo-rachidien (liquide dans lequel baigne le cerveau). Ces prélèvements sont effectués dans le cadre de la prise en charge standard et non pas spécifiquement pour le projet. Avec votre accord, ces prélèvements seront conservés et utilisés pour le projet.

Ces informations et prélèvements nous permettrons de chercher des facteurs communs susceptibles d'expliquer pourquoi certaines personnes sont plus à risques vis-à-vis des anévrismes que d'autres.

Le nombre de personnes recrutées aux Hôpitaux Universitaire Genevois pour ce projet sera d'environ 150 patient·e·s par an, 45 membres de la famille par an et 105 volontaires sain·e·s par an. A l'heure actuelle, il est prévu de conserver les informations et les échantillons pour une période initiale de 20 ans.

Ce projet est réalisé dans le respect des prescriptions de la législation Suisse. Nous suivons en outre l'ensemble des directives reconnues au niveau international. La commission d'éthique compétente a examiné et autorisé ce projet.

#### 3. Déroulement du projet

- Si vous acceptez de participer en tant que patient·e :
  - Des informations vous concernant et concernant votre anévrisme (scanners, IRM, radiographies et angiogrammes) seront relevées à partir de votre dossier hospitalier.




- O Des échantillons de sang seront prélevés. La prise de sang sera faite lors d'une visite de routine. Les échantillons de sang seront prélevés soit pour : A) l'étude génétique et l'analyse des modifications d'expression des gènes et des protéines dans le sang (3 échantillons de sang pour un volume maximal de 39 ml), soit B) pour l'étude bactériologique (3 échantillons de sang pour un volume maximal de 17 ml). Si votre anévrisme est traité, une prise de sang supplémentaire pourra être faite avant le traitement de votre anévrisme ou dans les 48 heures suivant le traitement de votre anévrisme et lors d'une visite de routine pour le contrôle de votre anévrisme (2 échantillons de sang pour un volume maximal de 22 ml pour l'analyse des modifications d'expression des gènes et des protéines dans le sang, ou, 3 échantillons de sang pour un volume maximal de 17 ml pour l'analyse bactériologique).
- Un échantillon de salive sera prélevé lors d'une visite de routine pour la surveillance de votre anévrisme, et/ou avant le traitement de votre anévrisme, et/ou après le traitement de votre anévrisme (6 mois après l'arrêt de tout traitement antibiotique).
- Un échantillon de selles sera prélevé lors d'une visite de routine pour la surveillance de votre anévrisme, et/ou avant le traitement de votre anévrisme, et/ou après le traitement de votre anévrisme (6 mois après l'arrêt de tout traitement antibiotique).
- Il vous sera demandé de compléter un questionnaire sur votre qualité de vie (durée d'environ 15 minutes). Ce questionnaire vous sera donné lors de votre première visite et lors de visites de routine effectuées pour le contrôle de votre anévrisme.
- Si votre anévrisme est traité, une partie de celui-ci pourra être prélevé, ainsi que du liquide céphalo-rachidien. Ces prélèvements sont effectués dans le cadre de la prise en charge standard et non pas spécifiquement pour le projet. Avec votre accord, ces prélèvements seront conservés et utilisés pour le projet.
- Vous pourriez aussi être contacté·e en dehors des visites de routine, soit pour vous demander des informations complémentaires, soit pour vous proposer de participer à d'autres études cliniques.
- Si vous acceptez de participer en tant que membre de la famille ou en tant que volontaire sain : e :
  - Des informations vous concernant seront relevées à partir de votre dossier hospitalier ou seront récoltées lors d'une visite avec la médecin-investigatrice/le médecin-investigateur ou un membre de son équipe.
  - Des échantillons de sang, de salive et/ou de selles seront prélevés. La prise de sang et la collecte de salive et de selles seront faits lors de la visite avec la médecin-investigatrice/le médecin-investigateur ou un membre de son équipe. Les échantillons de sang seront prélevés soit pour l'étude génétique et l'analyse des modifications d'expression des gènes et des protéines (3 échantillons de sang pour un volume maximal de 39 ml), soit pour l'étude bactériologique (3 échantillons de sang pour un volume maximal de 17 ml).
  - Il vous sera demandé de compléter un questionnaire sur votre qualité de vie (durée d'environ 15 minutes). Ce questionnaire vous sera donné lors de votre visite avec la médecininvestigatrice/le médecin-investigateur ou un membre de son équipe. Par envoi postal ou électronique, il vous sera demandé de remplir ce questionnaire sur votre qualité de vie environ tous les 5 ans.
  - Aucun examen radiologique ne sera effectué chez les membres de la famille et les volontaires sain·e·s spécifiquement pour ce projet. Aucune exigence n'est imposée, mais selon les recommandations internationales, il est recommandé aux membres de famille de patients atteints d'anévrismes cérébraux de réaliser un examen d'imagerie de dépistage pour les anévrismes cérébraux, examen pris en charge par les assurances maladies. Si cet examen est réalisé, les résultats seront intégrés à la base de données si la participante/le participant donne son accord.
  - Vous pourriez aussi être contacté·e en dehors de cette visite, soit pour vous demander des informations complémentaires, soit pour vous proposer de participer à d'autres études cliniques.




Il se peut que nous devions vous exclure du projet avant le terme prévu. Cette situation peut se produire si le projet est interrompu précocement et qu'il est demandé que les données soient détruites. Vous en seriez alors informé.e.

Avec votre accord, votre médecin traitant·e sera informé·e de votre participation au projet.

#### 4. Bénéfices

Votre participation au projet ne vous apportera aucun bénéfice.

Les résultats de ces recherches pourraient se révéler importants par la suite pour les personnes touchées par les anévrismes cérébraux.

# 5. Caractère facultatif de la participation et obligations

Votre participation est entièrement libre. Si vous choisissez de ne pas participer ou si vous choisissez de participer et revenez sur votre décision pendant le déroulement du projet, vous n'aurez pas à vous justifier. Cette décision n'aura pas de répercussions défavorables sur la suite de votre prise en charge médicale.

Si vous choisissez de participer à ce projet de recherche, vous serez tenu·e :

- de suivre les instructions et de remplir les exigences prévues par le protocole de recherche
   :
- d'informer la médecin-investigatrice/le médecin-investigateur de l'évolution de la maladie et de lui signaler tout nouveau symptôme, tout nouveau trouble et tout changement dans votre état :
- d'informer la médecin-investigatrice/le médecin-investigateur de tout traitement ou thérapie prescrit·e par une autre/un autre médecin ainsi que de tous les médicaments que vous prenez, même sans ordonnance.

## 6. Risques et contraintes

Les risques associés à cette étude sont ceux liés à la réalisation d'une ou plusieurs prises de sang (risque infectieux faible, hématome) et à l'utilisation d'un réseau informatique pour le transfert des données dont la sécurité ne peut jamais être totalement garantie.

Nous nous efforcerons de rendre les prises de sang aussi peu douloureuses que possible et mettrons en place des mesures de sécurité pour tous nos transferts de données codées.

Si certains résultats issus du projet (découverte de maladies lors des examens radiologiques ou sanguins) étaient susceptibles d'engendrer des inquiétudes chez vous, nous vous proposerons un soutien psychologique.

# 7. Alternatives

Si vous ne souhaitez pas participer à ce projet de recherche, mais vous restez ouvert à la possibilité d'une participation à d'autres projets, merci de l'indiquer à la médecin-investigatrice/au médecin-investigateur.

# 8. Résultats

Le projet permet d'obtenir différents résultats :

- 1. des résultats individuels qui vous concernent directement,
- 2. des résultats individuels découverts par hasard (ce qu'on appelle les découvertes fortuites),
- 3. les résultats définitifs objectifs du projet dans son ensemble.
- 1. La médecin-investigatrice/le médecin-investigateur vous avisera pendant le projet de toute nouvelle découverte importante vous concernant. Vous serez informé e oralement et par écrit ; vous pourrez par la suite à nouveau décider si vous souhaitez poursuivre votre participation au projet.




2. Les découvertes fortuites constituent des « résultats concomitants », à savoir des résultats qui n'ont pas été explicitement recherchés, mais qui ont été obtenus par hasard. Il peut s'agir p. ex. de résultats d'analyses génétiques ou de procédés d'imagerie.

Vous serez informé·e des découvertes fortuites si elles ont une incidence sur votre santé. Cela signifie que ces découvertes vous sont communiquées si l'on constate par hasard une pathologie qui n'était pas encore connue jusqu'alors ou que l'on peut empêcher l'apparition d'une maladie par des mesures de prévention. Si vous ne souhaitez pas recevoir ces informations (« droit de ne pas savoir »), merci de l'indiquer à la médecin-investigatrice/au médecin-investigateur.

Certains résultats pourraient nécessiter un test de confirmation. Une fois confirmés, ces résultats seront directement ajoutés à votre dossier médical et pourraient donc être consultés par toute personne à qui vous donnez accès à ce dossier (par exemple, un employeur ou une compagnie d'assurance).

3. La médecin-investigatrice/le médecin-investigateur peut vous faire parvenir, à l'issue du projet, une synthèse des résultats globaux.

## 9. Confidentialité des données et des échantillons

#### 9.1. Traitement et codage des données

Dans le cadre de ce projet de recherche, des données relatives à votre personne et à votre santé sont recueillies et traitées, en partie de manière automatisée. Ces informations sont codées au moment du relevé. Le codage signifie que toutes les données permettant de vous identifier (nom, date de naissance, etc.) sont remplacées par un code. Il n'est pas possible de relier les données à votre personne sans le code, qui reste en permanence au sein des Hôpitaux Universitaire de Genève. Seul un nombre limité de personnes peut consulter vos données sous une forme non codée, et ce, exclusivement afin de pouvoir accomplir des tâches nécessaires au déroulement du projet. Ces personnes sont tenues au secret professionnel. En tant que participant·e, vous avez à tout moment le droit de consulter vos données.

La base de données proprement dite sera également conservée après la fin de @neurIST et pourra être mise à disposition, sous forme codée, à d'autres chercheurs, éventuellement contre rémunération, voire développée dans le cadre d'applications commerciales.

## 9.2. Protection des données et des échantillons

Toutes les directives relatives à la protection des données sont rigoureusement respectées. Il est possible que vos données doivent être transmises sous forme codée, par exemple pour une publication, et qu'elles puissent être mises à la disposition d'autres chercheur·e·s.

Lorsque des données relatives à la santé ou des échantillons biologiques sont conservés sur place, ils constituent une banque de données ou une biobanque à des fins de recherche. Il se peut que ces données et ces échantillons soient envoyés sous forme codée dans le cadre de ce projet à une autre banque de données/biobanque. Vous pouvez demander la liste des institutions collaboratrices à la médecin investigatrice/au médecin investigateur.

Le promoteur doit s'assurer que le pays de destination garantit une protection des données équivalente à celle garantie en Suisse.

#### 9.3. Protection des données en cas de réutilisation

Vos données et échantillons pourraient ultérieurement se révéler importants pour répondre à d'autres questionnements et être envoyés à une autre banque de données/biobanque située en Suisse ou à l'étranger pour être aussi exploités dans d'autres projets de recherche (réutilisation). Cette banque de données/biobanque doit toutefois obéir aux mêmes normes et exigences que la banque de données/biobanque du présent projet.

Pour cette réutilisation, nous vous prions de signer le document prévu à cet effet (Déclaration de consentement pour la réutilisation de données et échantillons biologiques sous une forme codée). Ce deuxième consentement est indépendant de la participation au projet.




# 9.4. Protection des données en cas d'analyses génétiques

Dès lors que l'on procède à un relevé, un enregistrement ou une transmission de données issues de vos échantillons dans le cadre de la recherche génétique, il existe des risques liés à la confidentialité (p. ex., la possibilité de vous identifier), en particulier concernant les informations sur votre matériel génétique. Ces risques ne peuvent pas être totalement exclus et augmentent avec la quantité de données pouvant être appariées, notamment si vous publiez vous-même des données génétiques sur Internet (p. ex. à des fins de recherche généalogique). Les informations relatives à votre matériel génétique peuvent également être importantes pour les membres de votre famille ou votre planification familiale. Le promoteur prend toutes les mesures nécessaires pour réduire le plus possible les risques liés à la confidentialité.

# 9.5. Droit de consultation dans le cadre d'inspections

Le projet peut faire l'objet d'inspections. Celles-ci peuvent être effectuées par la commission d'éthique compétente ou par le promoteur qui a initié le projet. La médecin-investigatrice/le médecin-investigateur doit alors communiquer vos données pour les besoins de ces inspections. Toutes les personnes impliquées sont tenues au plus strict secret professionnel.

# 10. Retrait du projet

Vous pouvez à tout moment vous retirer du projet si vous le souhaitez. Vous n'avez pas à justifier vos décisions. Les données médicales recueillies jusque-là seront tout de même analysées car une fois intégrées à la base de données leur destruction devient impossible. Vous pourrez choisir sur la déclaration de retrait de consentement de l'étude @neurIST si vous souhaitez que :

- vos données soient gardées sous forme codée (codée signifie que votre matériel biologique et vos données ne peuvent être mis en relation avec votre personne qu'au moyen d'une clé) ou anonymisée (anonymisée signifie que le code reliant vos données à votre personne sera effacé, plus personne ne pourra savoir que ces données et ces échantillons sont les vôtres). Ce procédé vise avant tout à assurer la protection de données;
- o vos échantillons soient conservés ou détruits.

#### 11. Rémunération

Vous ne percevrez aucune rémunération pour votre participation à ce projet de recherche.

Les dépenses, telles que les frais de transport, qui découlent directement de la participation au projet vous seront remboursées.

Les prises de sang et les prélèvements de salive et de selles faits uniquement pour ce projet seront prises en charge par @neurIST.

Votre participation n'aura aucune conséquence financière pour vous ou votre assurance maladie.

Dans certains cas, les résultats de ce projet peuvent aider à développer des produits commerciaux. Si vous consentez à participer à ce projet, vous renoncez dans le même temps à tout droit d'exploitation commerciale (découlant de brevets en particulier).

# 12. Responsabilité

Les Hôpitaux Universitaire de Genève qui ont initié le projet de recherche et sont chargés de sa réalisation sont responsables des dommages que vous pourriez subir en relation avec le projet. Les conditions et la procédure sont fixées par la loi. Tous les actes étudiés dans cette étude font partie de la pratique quotidienne et relèvent de standards médicaux ne nécessitant pas une assurance spécifique à l'étude. La responsabilité civile de l'hôpital couvre les dommages éventuels imputables au projet que vous pourriez subir. Si vous subissiez un dommage du fait de votre participation au projet, il vous faudrait vous adresser au responsable du projet, le Dr Bijlenga.




## 13. Financement

Le projet est financé par des sources publiques pour l'exploitation académique des données. La coordination du financement est assurée par le bureau @neurIST de la Société européenne pour les traitements neurologiques minimalement invasifs ESMINT (www.esmint.eu). Il est actuellement financé par l'initiation continue de nouveaux projets déposés au Fonds National Suisse pour la recherche ainsi que dans d'autres organismes finançant la recherche en Europe.

# 14. Interlocuteur(s)

Vous pouvez à tout moment poser des questions au sujet du projet. En cas d'incertitudes pendant ou après le projet, vous pouvez vous adresser à :

Dr Philippe Bijlenga, responsable du projet : 079 204 40 43

Secrétariat du Dr Bijlenga : 022 372 34 26 En écrivant à aneurist : ccc@hcuge.ch

En consultant notre site internet : www.aneurist.org




## Déclaration de consentement

# Déclaration de consentement écrite pour la participation à un projet de recherche

Veuillez lire attentivement ce formulaire. N'hésitez pas à poser des questions lorsque vous ne comprenez pas quelque chose ou que vous souhaitez avoir des précisions. Votre consentement écrit est nécessaire pour participer au projet.

| Numéro BASEC du projet de recherche (après soumission à la commission d'éthique compétente) : | 2022-00426 |
|---|---|
| Titre<br>(scientifique et usuel) : | @neurIST : informatique biomédicale intégrée pour la gestion des anévrismes cérébraux |
| Institution responsable<br>(responsable du projet et adresse<br>complète) : | Hôpitaux Universitaire de Genève<br>Rue Micheli-du-Crest 24<br>1211 Genève 14 |
| Lieu de réalisation : | Genève, Suisse |
| Responsable du projet sur le site :<br>Nom et prénom en caractères d'imprimerie : | Dr Philippe Bijlenga |
| Participante / Participant :<br>Nom et prénom en caractères d'imprimerie :<br>Date de naissance : | |

- Je déclare avoir été informé·e, par la médecin-investigatrice/le médecin-investigateur soussigné·e, oralement et par écrit, des objectifs et du déroulement du projet de recherche ainsi que des avantages et des inconvénients possibles et des risques éventuels.
- Je prends part à ce projet de façon volontaire et j'accepte le contenu de la feuille d'information qui m'a été remise sur le projet précité. J'ai eu suffisamment de temps pour prendre ma décision.
- J'ai reçu les réponses aux questions que j'ai posées en relation avec la participation à ce projet.
   Je conserve la feuille d'information et reçois une copie de ma déclaration de consentement écrite.
- J'accepte que les spécialistes compétent·e·s de la direction de ce projet et de la commission d'éthique compétente puissent consulter mes données non codées afin de procéder à des contrôles et des inspections, à condition toutefois que la confidentialité de ces données soit strictement assurée.
- Je serai informé·e des résultats ayant une incidence directe sur ma santé. Si je ne souhaite pas obtenir ces informations, je prends contact avec la médecin-investigatrice/le médecin-investigateur.
- Si je bénéficie / devais bénéficier d'un traitement médical en dehors de l'institution responsable de ce projet, j'accepte que le médecin responsable du projet contacte ma/mon médecin traitant·e et que celui-ci lui fournisse des données médicales me concernant pouvant être pertinentes pour ce projet.
- Je sais que mes données personnelles, mes données de santé, et mes échantillons peuvent être transmis à des fins de recherche dans le cadre de ce projet et uniquement sous une forme codée. Le promoteur assure une protection des données conforme aux normes et exigences Suisses.
- Je peux, à tout moment et sans avoir à me justifier, révoquer mon consentement à participer au projet, sans que cette décision n'ait de répercussions défavorables sur la suite de ma prise en




charge. Les données et les échantillons recueillis jusqu'au retrait seront cependant analysés dans le cadre du projet.

- Je suis informé·e que les Hôpitaux Universitaire Genevois sont responsables des dommages éventuels imputables au projet.
- Je suis conscient e que les obligations mentionnées dans la feuille d'information destinée aux participant e s doivent être respectées pendant toute la durée du projet. La médecininvestigatrice/le médecin-investigateur peut m'exclure à tout moment du projet dans l'intérêt de ma santé.

| 0 | Je consens à participer à cette étude, j'accepte de donner accès à mon dossier de santé, qu'un lien soit créé entre ce dossier et la base de données locale @neurIST, et de remplir un questionnaire sur mon histoire clinique : Oui Non |
|---|---|
| 0 | J'accepte de fournir à @neurIST des données sous forme de clichés : Oui Non |
| 0 | J'accepte que des échantillons biologiques retirés dans un but thérapeutique soient étudiés : Oui Non |
| 0 | J'accepte de fournir des échantillons de sang selon le protocole : Oui Non |
| 0 | J'accepte de fournir des échantillons de salive selon le protocole : Oui Non |
| 0 | J'accepte de fournir des échantillons de selles selon le protocole : Oui Non |
| 0 | J'accepte d'être recontacté·e par @neurIST en vue d'autres consentements ou pour fournir de plus amples informations : Oui Non |
| 0 | Dans l'hypothèse où je ne pourrai pas être contacté·e pendant 3 mois, j'accepte que ma/mon médecin traitant·e puisse être contacté·e par un membre de l'équipe du projet afin d'obtenir de sa part des renseignements sur l'endroit où je me trouve ainsi que des informations médicales permettant de statuer sur l'évolution de l'affection cérébro-vasculaire : Oui Non |
| 0 | Je voudrais que ma/mon médecin traitant·e soit informé·e de ma participation à cette étude : Oui Non |




Veuillez étudier les points suivants avant de décider si vous souhaitez être informé·e des résultats de la recherche susceptibles d'être pertinents pour votre santé (ces résultats pourraient ne pas être disponibles avant 4 ans) :

- Ces résultats seront mis dans votre dossier médical.
- Ces résultats peuvent signaler l'existence d'un risque chez les personnes qui vous sont apparentées, et donc avoir des incidences sur votre famille.
- Vous devrez peut-être subir de nouveaux tests.
- Certains résultats pourraient évoquer des inquiétudes justifiant de recevoir un soutien psychologique.

| <ul> <li>Je souhaite être informérésultats susceptibles de m</li> <li>Oui</li> <li>Non</li> </ul> | e par la médecin-investigatrice/le médecin-investigateur des<br>e concerner : |
|---|---|
| Je souhaite que ma/mon m<br>concerner : Oui Non | édecin traitant·e soit informé·e des résultats susceptibles de me |
| Médecin Traitant·e : Nom, Prénom | |
| <u>Si pas de médecin traitant·e : autre</u> | e personne de contact : Nom, Prénom |
| Lieu, date | Signature de la participante/du participant |
| avoir expliqué à la participante/au p<br>satisfaire à toutes les obligations er<br>Si je devais prendre connaissance | tigatrice/du médecin-investigateur: Par la présente, j'atteste participant la nature, l'importance et la portée du projet. Je déclare n' relation avec ce projet conformément au droit suisse en vigueur. e, à quelque moment que ce soit durant la réalisation du projet, ur le consentement de la participante/du participant à prendre part ner immédiatement. |
| Lieu, date | Nom et prénom de la médecine-investigatrice/du médecin-<br>investigateur en caractères d'imprimerie. |
| | Signature de la médecine-investigatrice/du médecin-investigateur |




Demande de participation à un projet de recherche médical :

## @neurIST : informatique biomédicale intégrée pour la gestion des anévrismes cérébraux

#### Madame, Monsieur

Vous avez été intégré·e à un projet de recherche en situation d'urgence. Nous vous faisons parvenir le présent document pour vous informer de notre projet de recherche. Nous vous demandons de nous accorder, avec effet rétroactif, votre consentement pour la participation au projet.

Votre participation est entièrement libre. Toutes les données collectées dans le cadre de ce projet sont soumises à des règles strictes en matière de protection des données.

Le projet de recherche est mené par les Hôpitaux Universitaire de Genève. Nous vous en communiquerons les résultats si vous le souhaitez.

Lors d'un entretien, nous vous présenterons les éléments essentiels et répondrons à vos questions. Pour vous proposer d'ores et déjà un aperçu du projet, voici les points clés à retenir. Vous trouverez à la suite des informations complémentaires plus détaillées.

# Pourquoi menons-nous ce projet de recherche?

- Notre projet porte sur les anévrismes cérébraux qui sont des anomalies observées sur les vaisseaux sanguins irriguant notre cerveau. Les anévrismes cérébraux sont diagnostiqués par radiographie, scanners, angiographie ou IRM. Lors de la rupture d'un anévrisme cérébral, le traitement de cet anévrisme est indispensable pour permettre la survie de la patiente/du patient.
- Notre projet de recherche vise à déterminer les causes et les évolutions des anévrismes cérébraux afin d'améliorer leur prise en charge.
- La participation à ce projet est ouverte aux :
  - o Patient·e·s chez qui un anévrisme cérébral a été diagnostiqué ;
  - Membres d'une famille chez qui des personnes liées par le sang sont affectées par un anévrisme cérébral;
  - o Personnes ne souffrant pas d'anévrisme cérébral (Volontaire sain·e).

# Que dois-je faire si j'accepte de participer? – Que se passe-t-il pour moi en cas de participation?

- Forme de la participation : Si vous acceptez de participer à notre projet en tant que patient e diagnostiqué e avec un anévrisme cérébral, nous récolterons des informations générales vous concernant et nous vous prélèverons du sang, de la salive et des selles. Nous conserverons pour la recherche les tissus et le liquide enlevés dans le cadre du traitement de l'anévrisme.
- Déroulement pour les participant·e·s : la participation à cette étude implique, en plus de votre suivi habituel, une ou plusieurs prise·s de sang, le prélèvement de salive et de selles, et un questionnaire sur votre qualité de vie que vous devrez remplir lors de visites de routine. Des informations vous concernant et concernant votre anévrisme seront relevées à partir de votre dossier hospitalier. Vous pourrez aussi




être contacté·e pour fournir des informations complémentaires ou pour donner votre autorisation pour d'autres études cliniques

# Quels sont les bénéfices et les risques liés à la participation au projet ?

## Bénéfices

- Votre participation à ce projet de recherche ne vous apportera aucun bénéfice direct.
- Par votre participation, vous contribuez à aider les futur·e·s patient·e·s.

# Risques et contraintes

• Les risques associés à cette étude sont ceux liés à la réalisation d'une prise de sang (risque infectieux faible, hématome) et à l'utilisation d'un réseau informatique pour le transfert des données dont la sécurité ne peut jamais être totalement garantie.

En apposant votre signature à la fin du document, vous certifiez en avoir compris le contenu et consentir librement à prendre part au projet.




#### Information détaillée

## 1. Objectif du projet et sélection des participant·e·s

Dans cette feuille d'information, notre projet de recherche est aussi simplement désigné par le terme *projet*. Si vous acceptez d'y prendre part, vous êtes *un participant/une participante au projet*.

Ce projet permettra de mieux comprendre les causes et les évolutions des anévrismes cérébraux afin d'améliorer leur prise en charge. Ce projet conduira en effet à la création d'un système informatisé d'aide à la décision pour le traitement des anévrismes cérébraux.

Nous vous sollicitons car la participation est ouverte aux :

- o Patient·e·s chez qui un anévrisme cérébral a été diagnostiqué ;
- Membres d'une famille chez qui deux personnes liées par le sang sont affectées par un anévrisme cérébral;
- Aux personnes non diagnostiquées préalablement avec un anévrisme cérébral et dont deux membres de la famille non pas non plus été diagnostiqués préalablement avec un anévrisme cérébral, autrement dit toute personne ignorant avoir elle-même un antécédent d'anévrisme cérébral ou qu'un membre de sa famille lié par le sang ai un antécédent d'anévrisme cérébral : Volontaire sain e

# 2. Informations générales sur le projet

Ce projet international regroupant plusieurs centres hospitaliers a débuté en 2006. Les études menées sur les anévrismes cérébraux suggèrent que plusieurs facteurs sont impliqués dans l'apparition et l'évolution de cette maladie. Parmi ces facteurs, nos gènes, nos protéines et notre microbiote (bactéries vivant dans notre bouche et notre système digestif) semblent jouer un rôle important. Bien qu'il ait été montré que des modifications du microbiote par l'alimentation ou la consommation d'antibiotiques influence l'évolution de diverses maladies, son rôle dans l'apparition et l'évolution des anévrismes cérébraux n'est pas clairement défini.

Nous récolterons des informations générales vous concernant et nous vous prélèverons du sang, de la salive et des selles.

Nous récolterons également des informations concernant votre anévrisme. Lors de l'intervention pour le traitement de votre anévrisme, une partie de celui-ci a été prélevé, ainsi que du liquide céphalo-rachidien (liquide dans lequel baigne le cerveau). Ces prélèvements ont été effectués dans le cadre de la prise en charge standard et non pas spécifiquement pour le projet. Avec votre accord, ces prélèvements seront conservés et utilisés pour le projet.

Ces informations et prélèvements nous permettrons de chercher des facteurs communs susceptibles d'expliquer pourquoi certaines personnes sont plus à risques vis-à-vis des anévrismes que d'autres.

Le nombre de personnes recrutées aux Hôpitaux Universitaire Genevois pour ce projet sera d'environ 150 patient·e·s par an, 45 membres de la famille par an et 105 volontaires sain·e·s par an. A l'heure actuelle, il est prévu de conserver les informations et les échantillons pour une période initiale de 20 ans.

Ce projet est réalisé dans le respect des prescriptions de la législation Suisse. Nous suivons en outre l'ensemble des directives reconnues au niveau international. La commission d'éthique compétente a examiné et autorisé ce projet.

## 3. Déroulement du projet

- Si vous acceptez de participer :
  - o Des informations vous concernant et concernant votre anévrisme (scanners, IRM, radiographies et angiogrammes) seront relevées à partir de votre dossier hospitalier.
  - Des échantillons de sang seront prélevés. La prise de sang sera faite lors d'une visite de routine. Les échantillons de sang seront prélevés soit pour : A) l'étude génétique et l'analyse




des modifications d'expression des gènes et des protéines dans le sang (3 échantillons de sang pour un volume maximal de 39 ml), soit B) pour l'étude bactériologique (3 échantillons de sang pour un volume maximal de 17 ml). Lors du traitement de votre anévrisme, une prise de sang a été faite. Une autre pourra être faite dans les 48 heures suivant le traitement de votre anévrisme et lors d'une visite de routine (2 échantillons de sang pour un volume maximal de 22 ml pour l'analyse des modifications d'expression des gènes et des protéines dans le sang, ou, 3 échantillons de sang pour un volume maximal de 17 ml pour l'analyse bactériologique).

- Un échantillon de salive a été prélevé lors du traitement de votre anévrisme. Un autre échantillon sera prélevé lors d'une visite de routine après le traitement de l'anévrisme (6 mois après l'arrêt de tout traitement antibiotique).
- Un échantillon de selles a été prélevé lors du traitement de votre anévrisme. Un autre échantillon sera prélevé lors d'une visite de routine après le traitement de l'anévrisme (6 mois après l'arrêt de tout traitement antibiotique).
- Il vous sera demandé de compléter un questionnaire sur votre qualité de vie (durée d'environ 15 minutes). Ce questionnaire vous sera donné lors de votre première visite et lors de visites de routine effectuées pour le contrôle de votre anévrisme.
- Lors du traitement de votre anévrisme, une partie de celui-ci a été prélevé, ainsi que du liquide céphalo-rachidien. Ces prélèvements sont effectués dans le cadre de la prise en charge standard et non pas spécifiquement pour le projet. Avec votre accord, ces prélèvements seront conservés et utilisés pour le projet.
- Vous pourriez aussi être contacté·e en dehors des visites de routine, soit pour vous demander des informations complémentaires, soit pour vous proposer de participer à d'autres études cliniques.

Il se peut que nous devions vous exclure du projet avant le terme prévu. Cette situation peut se produire si le projet est interrompu précocement et qu'il est demandé que les données soient détruites. Vous en seriez alors informé·e.

Avec votre accord, votre médecin traitant·e sera informé·e de votre participation au projet.

#### 4. Bénéfices

Votre participation au projet ne vous apportera aucun bénéfice.

Les résultats de ces recherches pourraient se révéler importants par la suite pour les personnes touchées par les anévrismes cérébraux.

## 5. Caractère facultatif de la participation et obligations

Votre participation est entièrement libre. Si vous choisissez de ne pas participer ou si vous choisissez de participer et revenez sur votre décision pendant le déroulement du projet, vous n'aurez pas à vous justifier. Cette décision n'aura pas de répercussions défavorables sur la suite de votre prise en charge médicale.

Si vous choisissez de participer à ce projet de recherche, vous serez tenu·e:

- o de suivre les instructions et de remplir les exigences prévues par le protocole de recherche;
- d'informer la médecin-investigatrice/le médecin-investigateur de l'évolution de la maladie et de lui signaler tout nouveau symptôme, tout nouveau trouble et tout changement dans votre état;
- o d'informer la médecin-investigatrice/le médecin-investigateur de tout traitement ou thérapie prescrit·e par une autre/un autre médecin ainsi que de tous les médicaments que vous prenez, même sans ordonnance.

## 6. Risques et contraintes

Les risques associés à cette étude sont ceux liés à la réalisation d'une ou plusieurs prises de sang (risque infectieux faible, hématome) et à l'utilisation d'un réseau informatique pour le transfert des données dont la sécurité ne peut jamais être totalement garantie.




Nous nous efforcerons de rendre les prises de sang aussi peu douloureuses que possible et mettrons en place des mesures de sécurité pour tous nos transferts de données codées.

Si certains résultats issus du projet (découverte de maladies lors des examens radiologiques ou sanguins) étaient susceptibles d'engendrer des inquiétudes chez vous, nous vous proposerons un soutien psychologique.

#### 7. Alternatives

Si vous ne souhaitez pas participer à ce projet de recherche, mais vous restez ouvert à la possibilité d'une participation à d'autres projets, merci de l'indiquer à la médecin-investigatrice/au médecin-investigateur.

## 8. Résultats

Le projet permet d'obtenir différents résultats :

- 1. des résultats individuels qui vous concernent directement,
- 2. des résultats individuels découverts par hasard (ce qu'on appelle les découvertes fortuites).
- 3. les résultats définitifs objectifs du projet dans son ensemble.
- 1. La médecin-investigatrice/le médecin-investigateur vous avisera pendant le projet de toute nouvelle découverte importante vous concernant. Vous serez informé e oralement et par écrit ; vous pourrez par la suite à nouveau décider si vous souhaitez poursuivre votre participation au projet.
- 2. Les découvertes fortuites constituent des « résultats concomitants », à savoir des résultats qui n'ont pas été explicitement recherchés, mais qui ont été obtenus par hasard. Il peut s'agir p. ex. de résultats d'analyses génétiques ou de procédés d'imagerie.

Vous serez informé e des découvertes fortuites si elles ont une incidence sur votre santé. Cela signifie que ces découvertes vous sont communiquées si l'on constate par hasard une pathologie qui n'était pas encore connue jusqu'alors ou que l'on peut empêcher l'apparition d'une maladie par des mesures de prévention. Si vous ne souhaitez pas recevoir ces informations (« droit de ne pas savoir »), merci de l'indiquer à la médecin-investigatrice/au médecin-investigateur.

Certains résultats pourraient nécessiter un test de confirmation. Une fois confirmés, ces résultats seront directement ajoutés à votre dossier médical et pourraient donc être consultés par toute personne à qui vous donnez accès à ce dossier (par exemple, un employeur ou une compagnie d'assurance).

3. La médecin-investigatrice/le médecin-investigateur peut vous faire parvenir, à l'issue du projet, une synthèse des résultats globaux.

# 9. Confidentialité des données et des échantillons

# 9.1. Traitement et codage des données

Dans le cadre de ce projet de recherche, des données relatives à votre personne et à votre santé sont recueillies et traitées, en partie de manière automatisée. Ces informations sont codées au moment du relevé. Le codage signifie que toutes les données permettant de vous identifier (nom, date de naissance, etc.) sont remplacées par un code. Il n'est pas possible de relier les données à votre personne sans le code, qui reste en permanence au sein des Hôpitaux Universitaire de Genève. Seul un nombre limité de personnes peut consulter vos données sous une forme non codée, et ce, exclusivement afin de pouvoir accomplir des tâches nécessaires au déroulement du projet. Ces personnes sont tenues au secret professionnel. En tant que participant·e, vous avez à tout moment le droit de consulter vos données.

La base de données proprement dite sera également conservée après la fin de @neurIST et pourra être mise à disposition, sous forme codée, à d'autres chercheurs, éventuellement contre rémunération, voire développée dans le cadre d'applications commerciales.




#### 9.2. Protection des données et des échantillons

Toutes les directives relatives à la protection des données sont rigoureusement respectées. Il est possible que vos données doivent être transmises sous forme codée, par exemple pour une publication, et qu'elles puissent être mises à la disposition d'autres chercheur·e·s.

Lorsque des données relatives à la santé ou des échantillons biologiques sont conservés sur place, ils constituent une banque de données ou une biobanque à des fins de recherche. Il se peut que ces données et ces échantillons soient envoyés sous forme codée dans le cadre de ce projet à une autre banque de données/biobanque. Vous pouvez demander la liste des institutions collaboratrices à la médecin investigatrice/au médecin investigateur.

Le promoteur doit s'assurer que le pays de destination garantit une protection des données équivalente à celle garantie en Suisse.

#### 9.3. Protection des données en cas de réutilisation

Vos données et échantillons pourraient ultérieurement se révéler importants pour répondre à d'autres questionnements et être envoyés à une autre banque de données/biobanque située en Suisse ou à l'étranger pour être aussi exploités dans d'autres projets de recherche (réutilisation). Cette banque de données/biobanque doit toutefois obéir aux mêmes normes et exigences que la banque de données/biobanque du présent projet.

Pour cette réutilisation, nous vous prions de signer le document prévu à cet effet (Déclaration de consentement pour la réutilisation de données et échantillons biologiques sous une forme codée). Ce deuxième consentement est indépendant de la participation au projet.

# 9.4. Protection des données en cas d'analyses génétiques

Dès lors que l'on procède à un relevé, un enregistrement ou une transmission de données issues de vos échantillons dans le cadre de la recherche génétique, il existe des risques liés à la confidentialité (p. ex., la possibilité de vous identifier), en particulier concernant les informations sur votre matériel génétique. Ces risques ne peuvent pas être totalement exclus et augmentent avec la quantité de données pouvant être appariées, notamment si vous publiez vous-même des données génétiques sur Internet (p. ex. à des fins de recherche généalogique). Les informations relatives à votre matériel génétique peuvent également être importantes pour les membres de votre famille ou votre planification familiale. Le promoteur prend toutes les mesures nécessaires pour réduire le plus possible les risques liés à la confidentialité.

## 9.5. Droit de consultation dans le cadre d'inspections

Le projet peut faire l'objet d'inspections. Celles-ci peuvent être effectuées par la commission d'éthique compétente ou par le promoteur qui a initié le projet. La médecin-investigatrice/le médecin-investigateur doit alors communiquer vos données pour les besoins de ces inspections. Toutes les personnes impliquées sont tenues au plus strict secret professionnel.

# 10. Retrait du projet

Vous pouvez à tout moment vous retirer du projet si vous le souhaitez. Vous n'avez pas à justifier vos décisions. Les données médicales recueillies jusque-là seront tout de même analysées car une fois intégrées à la base de données leur destruction devient impossible. Vous pourrez choisir sur la déclaration de retrait de consentement de l'étude @neurIST si vous souhaitez que :

- vos données soient gardées sous forme codée (codée signifie que votre matériel biologique et vos données ne peuvent être mis en relation avec votre personne qu'au moyen d'une clé) ou anonymisée (anonymisée signifie que le code reliant vos données à votre personne sera effacé, plus personne ne pourra savoir que ces données et ces échantillons sont les vôtres). Ce procédé vise avant tout à assurer la protection de données :
- o vos échantillons soient conservés ou détruits.

# 11. Rémunération

Vous ne percevrez aucune rémunération pour votre participation à ce projet de recherche.




Les dépenses, telles que les frais de transport, qui découlent directement de la participation au projet vous seront remboursées.

Les prises de sang et les prélèvements de salive et de selles faits uniquement pour ce projet seront prises en charge par @neurIST.

Votre participation n'aura aucune conséquence financière pour vous ou votre assurance maladie.

Dans certains cas, les résultats de ce projet peuvent aider à développer des produits commerciaux. Si vous consentez à participer à ce projet, vous renoncez dans le même temps à tout droit d'exploitation commerciale (découlant de brevets en particulier).

## 12. Responsabilité

Les Hôpitaux Universitaire de Genève qui ont initié le projet de recherche et sont chargés de sa réalisation sont responsables des dommages que vous pourriez subir en relation avec le projet. Les conditions et la procédure sont fixées par la loi. Tous les actes étudiés dans cette étude font partie de la pratique quotidienne et relèvent de standards médicaux ne nécessitant pas une assurance spécifique à l'étude. La responsabilité civile de l'hôpital couvre les dommages éventuels imputables au projet que vous pourriez subir. Si vous subissiez un dommage du fait de votre participation au projet, il vous faudrait vous adresser au responsable du projet, le Dr Bijlenga.

#### 13. Financement

Le projet est financé par des sources publiques pour l'exploitation académique des données. La coordination du financement est assurée par le bureau @neurIST de la Société européenne pour les traitements neurologiques minimalement invasifs ESMINT (www.esmint.eu). Il est actuellement financé par l'initiation continue de nouveaux projets déposés au Fonds National Suisse pour la recherche ainsi que dans d'autres organismes finançant la recherche en Europe.

# 14. Interlocuteur(s)

Vous pouvez à tout moment poser des questions au sujet du projet. En cas d'incertitudes pendant ou après le projet, vous pouvez vous adresser à :

Dr Philippe Bijlenga, responsable du projet : 079 204 40 43

Secrétariat du Dr Bijlenga : 022 372 34 26 En écrivant à aneurist : ccc@hcuge.ch

En consultant notre site internet : www.aneurist.org




## Déclaration de consentement

# Déclaration de consentement écrite pour la participation à un projet de recherche

Veuillez lire attentivement ce formulaire. N'hésitez pas à poser des questions lorsque vous ne comprenez pas quelque chose ou que vous souhaitez avoir des précisions. Votre consentement écrit est nécessaire pour participer au projet.

| Numéro BASEC du projet de recherche<br>(après soumission à la commission<br>d'éthique compétente) : | 2022-00426 |
|---|---|
| Titre<br>(scientifique et usuel) : | @neurIST : informatique biomédicale intégrée pour la gestion des anévrismes cérébraux |
| Institution responsable<br>(responsable du projet et adresse<br>complète) : | Hôpitaux Universitaire de Genève<br>Rue Micheli-du-Crest 24<br>1211 Genève 14 |
| Lieu de réalisation : | Genève, Suisse |
| Responsable du projet sur le site :<br>Nom et prénom en caractères d'imprimerie : | Dr Philippe Bijlenga |
| Participante / Participant :<br>Nom et prénom en caractères d'imprimerie :<br>Date de naissance : | |

- Je déclare avoir été informé·e, par la médecin-investigatrice/le médecin-investigateur soussigné·e, oralement et par écrit, des objectifs et du déroulement du projet de recherche ainsi que des avantages et des inconvénients possibles et des risques éventuels.
- Je prends part à ce projet de façon volontaire et j'accepte le contenu de la feuille d'information qui m'a été remise sur le projet précité. J'ai eu suffisamment de temps pour prendre ma décision.
- J'ai reçu les réponses aux questions que j'ai posées en relation avec la participation à ce projet.
   Je conserve la feuille d'information et reçois une copie de ma déclaration de consentement écrite.
- J'accepte que les spécialistes compétent·e·s de la direction de ce projet et de la commission d'éthique compétente puissent consulter mes données non codées afin de procéder à des contrôles et des inspections, à condition toutefois que la confidentialité de ces données soit strictement assurée.
- Je serai informé·e des résultats ayant une incidence directe sur ma santé. Si je ne souhaite pas obtenir ces informations, je prends contact avec la médecin-investigatrice/le médecininvestigateur.
- Si je bénéficie / devais bénéficier d'un traitement médical en dehors de l'institution responsable de ce projet, j'accepte que le médecin responsable du projet contacte ma/mon médecin traitant·e et que celui-ci lui fournisse des données médicales me concernant pouvant être pertinentes pour ce projet.
- Je sais que mes données personnelles, mes données de santé, et mes échantillons peuvent être transmis à des fins de recherche dans le cadre de ce projet et uniquement sous une forme codée. Le promoteur assure une protection des données conforme aux normes et exigences Suisses.
- Je peux, à tout moment et sans avoir à me justifier, révoquer mon consentement à participer au projet, sans que cette décision n'ait de répercussions défavorables sur la suite de ma prise en




charge. Les données et les échantillons recueillis jusqu'au retrait seront cependant analysés dans le cadre du projet.

- Je suis informé·e que les Hôpitaux Universitaire Genevois sont responsables des dommages éventuels imputables au projet.
- Je suis conscient e que les obligations mentionnées dans la feuille d'information destinée aux participant e s doivent être respectées pendant toute la durée du projet. La médecininvestigatrice/le médecin-investigateur peut m'exclure à tout moment du projet dans l'intérêt de ma santé.

| 0 | Je consens à participer à cette étude, j'accepte de donner accès à mon dossier de santé, qu'un lien soit créé entre ce dossier et la base de données locale @neurIST, et de remplir un questionnaire sur mon histoire clinique : Oui Non |
|---|---|
| 0 | J'accepte de fournir à @neurIST des données sous forme de clichés : Oui Non |
| 0 | J'accepte que des échantillons biologiques retirés dans un but thérapeutique soient étudiés : Oui Non |
| 0 | J'accepte de fournir des échantillons de sang selon le protocole : Oui Non |
| 0 | J'accepte de fournir des échantillons de salive selon le protocole : Oui Non |
| 0 | J'accepte de fournir des échantillons de selles selon le protocole : Oui Non |
| 0 | J'accepte d'être recontacté·e par @neurIST en vue d'autres consentements ou pour fournir de plus amples informations : ☐ Oui ☐ Non |
| 0 | Dans l'hypothèse où je ne pourrai pas être contacté·e pendant 3 mois, j'accepte que ma/mon médecin traitant·e puisse être contacté·e par un membre de l'équipe du projet afin d'obtenir de sa part des renseignements sur l'endroit où je me trouve ainsi que des informations médicales permettant de statuer sur l'évolution de l'affection cérébro-vasculaire : Oui Non |
| 0 | Je voudrais que ma/mon médecin traitant·e soit informé·e de ma participation à cette étude : Oui Non |




Veuillez étudier les points suivants avant de décider si vous souhaitez être informé·e des résultats de la recherche susceptibles d'être pertinents pour votre santé (ces résultats pourraient ne pas être disponibles avant 4 ans) :

- Ces résultats seront mis dans votre dossier médical.
- Ces résultats peuvent signaler l'existence d'un risque chez les personnes qui vous sont apparentées, et donc avoir des incidences sur votre famille.
- Vous devrez peut-être subir de nouveaux tests.
- Certains résultats pourraient évoquer des inquiétudes justifiant de recevoir un soutien psychologique.

| <ul> <li>Je souhaite être informérésultats susceptibles de m</li> <li>Oui</li> <li>Non</li> </ul> | e par la médecin-investigatrice/le médecin-investigateur des<br>e concerner : |
|---|---|
| Je souhaite que ma/mon m<br>concerner : Oui Non | édecin traitant·e soit informé·e des résultats susceptibles de me |
| Médecin Traitant·e : Nom, Prénom | |
| <u>Si pas de médecin traitant·e : autre</u> | e personne de contact : Nom, Prénom |
| Lieu, date | Signature de la participante/du participant |
| avoir expliqué à la participante/au p<br>satisfaire à toutes les obligations er<br>Si je devais prendre connaissance | tigatrice/du médecin-investigateur: Par la présente, j'atteste participant la nature, l'importance et la portée du projet. Je déclare n' relation avec ce projet conformément au droit suisse en vigueur. e, à quelque moment que ce soit durant la réalisation du projet, ur le consentement de la participante/du participant à prendre part ner immédiatement. |
| Lieu, date | Nom et prénom de la médecine-investigatrice/du médecin-<br>investigateur en caractères d'imprimerie. |
| | Signature de la médecine-investigatrice/du médecin-investigateur |




# Confirmation écrite d'un médecin non associé au projet de recherche

Confirmation écrite pour le médecin non associé au projet de recherche, qui *n'*est *pas* impliqué dans le projet de recherche mentionné ci-après et qui défend les intérêts de la personne se prêtant à l'expérience (LRH art 30).

# Données sur le projet de recherche

| Titre du projet de recherche: @neurIST : informatique biomédicale intégrée pour la gestion des anévrismes cérébraux |
|---|
| Numéro du projet de recherche: |
| Lieu où se déroule le projet de recherche : Hôpitaux Universitaire de Genève |
| Nom et prénom du médecin investigateur responsable: Bijlenga Philippe |
| Nom et prénom du / de la participant·e: |
| Date de naissance (facultatif): sexe (facultatif): |

J'ai reçu et j'ai lu le résumé du protocole du projet de recherche susmentionné.

J'atteste que les intérêts du / de la participant ∙e sont respectés et que son suivi médical est garanti.

| nature du médecin non<br>ocié au projet de<br>nerche |
|------------------------------------------------------|
|------------------------------------------------------|

Par la présente, j'atteste avoir expliqué au médecin non associé au projet de recherche la nature, l'importance et la portée du projet. Si je devrai prendre connaissance, à quelque moment que ce soit durant la réalisation du projet, d'éléments susceptibles d'influer sur le consentement du / de la participant e à prendre part au projet de recherche, je m'engage à l'en informer immédiatement.

| Lieu, date | Nom, prénom et numéro de téléphone<br>de l'investigateur responsable (en<br>caractères d'imprimerie) | Signature de l'investigateur responsable |
|---|---|---|






Demande de participation à un projet de recherche médical :

# @neurIST : informatique biomédicale intégrée pour la gestion des anévrismes cérébraux

Madame, Monsieur,

Par la présente, nous souhaiterions vous informer de notre projet de recherche. La patiente/le patient, la personne placée sous votre responsabilité est incapable de discernement et, par-là, de communiquer sa volonté. Par conséquent, nous vous faisons parvenir la présente feuille d'information, qui vous permettra de vérifier si vous acceptez de faire participer la personne que vous représentez. En effet, vous pouvez accorder votre consentement en qualité de proche ou de représentant·e légal·e.

Ci-après, nous vous présentons le projet : d'abord, par un résumé pour vous donner un rapide aperçu ; puis par une description plus détaillée.




Demande de participation à un projet de recherche médical :

# @neurIST : informatique biomédicale intégrée pour la gestion des anévrismes cérébraux

Madame, Monsieur,

Nous vous proposons ici de nous accorder votre consentement pour la participation de la patiente/du patient à notre projet.

La participation est entièrement libre. Toutes les données collectées dans le cadre de ce projet sont soumises à des règles strictes en matière de protection des données.

Le projet de recherche est mené par les Hôpitaux Universitaire de Genève. Nous vous en communiquerons les résultats si vous le souhaitez.

Lors d'un entretien, nous vous présenterons les éléments essentiels et répondrons à vos questions. Pour vous proposer d'ores et déjà un aperçu du projet, voici les points clés à retenir. Vous trouverez à la suite des informations complémentaires plus détaillées.

# Pourquoi menons-nous ce projet de recherche?

- Notre projet porte sur les anévrismes cérébraux qui sont des anomalies observées sur les vaisseaux sanguins irriguant notre cerveau. Les anévrismes cérébraux sont diagnostiqués par radiographie, scanners, angiographie ou IRM. Lors de la rupture d'un anévrisme cérébral, le traitement de cet anévrisme est indispensable pour permettre la survie de la patiente/du patient.
- Notre projet de recherche vise à déterminer les causes et les évolutions des anévrismes cérébraux afin d'améliorer leur prise en charge.

# Que doit faire le patient en cas de participation ? – Que se passe-t-il pour le patient en cas de participation ?

- Forme de la participation: Si vous nous accordez votre consentement pour la participation de la patiente/du patient, nous récolterons des informations générales concernant la patiente/le patient et nous lui prélèverons du sang, de la salive et des selles. Nous conserverons pour la recherche les tissus et le liquide enlevés dans le cadre du traitement de l'anévrisme.
- Déroulement pour les participant·e·s: Si le patient participe au projet, sa participation à cette étude implique, en plus de son suivi habituel, une ou plusieurs prise(s) de sang, le prélèvement de salive et de selles, et un questionnaire sur sa qualité de vie qu'elle/il devra remplir lors de visites de routine. Des informations la/le concernant et concernant son anévrisme seront relevées à partir de son dossier hospitalier. La patiente/le patient pourra aussi être contacté pour fournir des informations complémentaires ou pour donner son autorisation pour d'autres études cliniques.




# Quels sont les bénéfices et les risques liés à la participation au projet ?

# Bénéfices pour les participants

- La participation à ce projet de recherche n'apportera à la patiente/au patient aucun bénéfice direct.
- Par sa participation, la patiente/le patient contribue à aider les futurs patient e.s.

# Risques et contraintes

 Les risques associés à cette étude sont ceux liés à la réalisation d'une prise de sang (risque infectieux faible, hématome) et à l'utilisation d'un réseau informatique pour le transfert des données dont la sécurité ne peut jamais être totalement garantie.

En apposant votre signature à la fin du document, vous attestez en avoir compris tout le contenu et accorder librement votre consentement pour la participation de la patiente/du patient au projet.




## Information détaillée

# 1. Objectif du projet et sélection des participant·e·s

Dans cette feuille d'information, notre projet de recherche est aussi simplement désigné par le terme *projet*. Si vous accordez votre consentement, en votre qualité de proche ou de représentant e légal e, pour la participation du patient, ce dernier est un e participant e au projet.

Ce projet permettra de mieux comprendre les causes et les évolutions des anévrismes cérébraux afin d'améliorer leur prise en charge. Ce projet conduira en effet à la création d'un système informatisé d'aide à la décision pour le traitement des anévrismes cérébraux.

Nous vous sollicitons en votre qualité de proche ou de représentant e légale, car la participation est ouverte à toutes les personnes chez qui un anévrisme cérébral a été diagnostiqué.

# 2. Informations générales sur le projet

Ce projet international regroupant plusieurs centres hospitaliers a débuté en 2006. Les études menées sur les anévrismes cérébraux suggèrent que plusieurs facteurs sont impliqués dans l'apparition et l'évolution de cette maladie. Parmi ces facteurs, nos gènes, nos protéines et notre microbiote (bactéries vivant dans notre bouche et notre système digestif) semblent jouer un rôle important. Bien qu'il ait été montré que des modifications du microbiote par l'alimentation ou la consommation d'antibiotiques influence l'évolution de diverses maladies, son rôle dans l'apparition et l'évolution des anévrismes cérébraux n'est pas clairement défini.

Nous récolterons des informations générales concernant tous les participant·e·s et nous prélèverons du sang, de la salive et des selles.

Nous récolterons également des informations concernant l'anévrisme de la patiente/du patient. Lors de l'intervention pour le traitement de l'anévrisme, une partie de celui-ci pourra être prélevé, ainsi que du liquide céphalo-rachidien (liquide dans lequel baigne le cerveau). Ces prélèvements sont effectués dans le cadre de la prise en charge standard et non pas spécifiquement pour le projet. Avec votre accord, ces prélèvements seront conservés pour le projet.

Ces informations et prélèvements nous permettrons de chercher des facteurs communs susceptibles d'expliquer pourquoi certaines personnes sont plus à risque vis-à-vis des anévrismes que d'autres.

Le nombre de personnes recrutées au HUG pour ce projet sera d'environ 150 patient·e·s par an, 45 membres de la famille par an et 105 volontaires sain·e·s par an. A l'heure actuelle, il est prévu de conserver les informations et les échantillons pour une période initiale de 20 ans.

Ce projet est réalisé dans le respect des prescriptions de la législation Suisse. Nous suivons en outre l'ensemble des directives reconnues au niveau international. La commission d'éthique compétente a examiné et autorisé ce projet.

# 3. Déroulement pour les participant·e·s

- Des informations concernant la patiente/le patient et concernant son anévrisme (scanners, IRM, radiographies et angiogrammes) seront relevées à partir de son dossier hospitalier.
- Des échantillons de sang seront prélevés. La prise de sang sera faite lors d'une visite de routine. Les échantillons de sang seront prélevés soit pour : A) l'étude génétique et l'analyse des modifications d'expression des gènes et des protéines dans le sang (3 échantillons de sang pour un volume maximal de 39 ml), soit B) pour l'étude bactériologique (3 échantillons de sang pour un volume maximal de 17 ml). Si l'anévrisme est traité, une prise de sang supplémentaire pourra être faite avant le traitement de l'anévrisme ou dans les 48 heures suivant le traitement de l'anévrisme et lors d'une visite de routine pour le contrôle de l'anévrisme (2 échantillons de sang pour un volume maximal de 22 ml pour l'analyse des modifications d'expression des gènes et des protéines dans le sang, ou, 3 échantillons de sang pour un volume maximal de 17 ml pour l'analyse bactériologique).




- Un échantillon de salive sera prélevé lors d'une visite de routine pour la surveillance de l'anévrisme, et/ou avant le traitement de l'anévrisme, et/ou après le traitement de l'anévrisme (6 mois après l'arrêt de tout traitement antibiotique).
- Un échantillon de selles sera prélevé lors d'une visite de routine pour la surveillance de l'anévrisme, et/ou avant le traitement de l'anévrisme, et/ou après le traitement de l'anévrisme (6 mois après l'arrêt de tout traitement antibiotique).
- Il sera demandé à la patiente/au patient de compléter, avec assistance (pour s'assurer de la compréhension), un questionnaire sur sa qualité de vie (durée d'environ 30 minutes). Ce questionnaire lui sera donné lors de sa première visite et lors des visites de routine effectuées pour le contrôle de son anévrisme.
- Si l'anévrisme de la patiente/du patient est traité, une partie de celui-ci pourra être prélevé, ainsi que du liquide céphalo-rachidien. Ces prélèvements sont effectués dans le cadre de la prise en charge standard et non pas spécifiquement pour le projet. Avec votre accord, ces prélèvements seront conservés pour le projet.
- Vous pourrez aussi être contacté·e en dehors des visites de routine de la patiente/du patient, soit pour vous demander des informations complémentaires, soit pour vous proposer que la patiente/le patient participe à d'autres études cliniques.

Il se peut que nous devions retirer la patiente/le patient du projet avant le terme prévu. Cette situation peut se produire si le projet est interrompu précocement et qu'il est demandé que les données soient détruites.

Avec votre accord, la médecin traitante/le médecin traitant sera informé de la participation de la patiente/du patient à ce projet.

# 4. Bénéfices pour les participant·e·s

La participation à ce projet de recherche n'apportera pas de bénéfice personnel à la patiente/au patient.

Les résultats des recherches pourraient se révéler importants par la suite pour les personnes touchées par la même maladie.

#### 5. Caractère facultatif de la participation et obligations

La participation au projet de recherche est entièrement libre. Si la patiente/le patient ne souhaite pas participer ou si vous, en tant que proche ou représentant e légal e, revenez ultérieurement sur votre décision à ce sujet, vous n'aurez pas à vous justifier. Cette décision n'aura pas de répercussions défavorables sur la suite de sa prise en charge médicale.

La participation au projet implique les obligations suivantes :

- la patiente/le patient est tenu·e de suivre les instructions et de remplir les exigences prévues par le protocole de recherche ;
- la médecin investigatrice/le médecin-investigateur doit être informé·e de l'évolution de la maladie et il convient de lui signaler tout nouveau symptôme, tout nouveau trouble et tout changement dans l'état de la patiente/du patient ;
- la médecin investigatrice/le médecin-investigateur doit être informé·e de tout traitement ou thérapie prescrit par un·e autre médecin ainsi que de tous les médicaments pris par la patiente/le patient, même sans ordonnance.

# 6. Risques et contraintes pour les participant·e·s

En participant au projet, la patiente/le patient ne sera exposé·e qu'à des risques mineurs tels qu'une prise de sang (risque infectieux faible, hématome) et à l'utilisation d'un réseau informatique pour le transfert des données dont la sécurité ne peut jamais être totalement garantie.

Nous nous efforcerons de rendre les prises de sang aussi peu douloureuses que possible et mettrons en place des mesures de sécurité pour tous nos transferts de données codées.

Si certains résultats issus du projet (découverte de maladies lors des examens radiologiques ou sanguins) étaient susceptibles d'engendrer des inquiétudes chez la patiente/le patient, nous lui proposerons un soutien psychologique.




#### 7. Alternatives

Si vous ne souhaitez pas que la patiente/le patient participe à ce projet de recherche, mais vous restez ouvert à la possibilité d'une participation à d'autres projets, merci de l'indiquer informer la médecin-investigatrice/le médecin-investigateur.

#### 8. Résultats

Le projet permet d'obtenir différents résultats :

- 1. des résultats individuels qui concernent directement la patiente/le patient,
- 2. des résultats individuels découverts par hasard (ce qu'on appelle les découvertes fortuites),
- 3. les résultats définitifs objectifs du projet dans son ensemble.
- 1. Au cours du projet, la médecin-investigatrice/le médecin-investigateur vous avisera, en votre qualité de proche ou de représentant·e légal·e, de toute nouvelle découverte importante pour la patiente/le patient. Vous serez informé·e oralement et par écrit ; vous pourrez par la suite à nouveau décider si la patiente/le patient doit poursuivre sa participation au projet.
- 2. Les découvertes fortuites constituent des « résultats concomitants », à savoir des résultats qui n'ont pas été explicitement recherchés, mais qui ont été obtenus par hasard. Il peut s'agir p. ex. de résultats d'analyses génétiques ou de procédés d'imagerie.

Vous serez informé·e des découvertes fortuites si elles ont une incidence sur la santé de la patiente/du patient. Cela signifie que ces découvertes sont communiquées si l'on constate par hasard une pathologie qui n'était pas encore connue jusqu'alors ou que l'on peut empêcher l'apparition d'une maladie par des mesures de prévention. Si vous ne souhaitez pas recevoir ces informations (« droit de ne pas savoir »), merci de l'indiquer à la médecin-investigatrice/au médecin-investigateur.

Certains résultats pourraient nécessiter un test de confirmation. Une fois confirmés, ces résultats seront directement ajoutés au dossier médical de la patiente/du patient et pourraient donc être consultés par toute personne à qui la patiente/le patient a donné accès au dossier (par exemple, un employeur ou une compagnie d'assurance).

3. La médecin-investigatrice/le médecin-investigateur peut vous faire parvenir, à l'issue du projet, une synthèse des résultats globaux.

# 9. Confidentialité des données et des échantillons

# 9.1. Traitement et codage des données

Dans le cadre de ce projet de recherche, des données relatives à la santé de la patiente/du patient sont recueillies et traitées, en partie de manière automatisée. Ces informations sont codées au moment du relevé. Le codage signifie que toutes les données permettant d'identifier la patiente/le patient (nom, date de naissance, etc.) sont effacées et remplacées par un code. Il n'est pas possible de relier les données à la patiente/au patient sans le code, qui reste en permanence au sein des Hôpitaux Universitaire de Genève.

Seul un nombre limité de personnes peut consulter les données de la patiente/du patient sous une forme non codée, et ce, exclusivement pour pouvoir accomplir les tâches nécessaires au déroulement du projet de recherche. Ces personnes sont tenues au secret professionnel. En votre qualité de proche ou représentant·e légal·e, vous avez le droit de consulter les données de la patiente/du patient.

La base de données proprement dite sera également conservée après la fin de @neurlST et pourra être mise à disposition, sous forme codée, à d'autres chercheurs, éventuellement contre rémunération, voire développée dans le cadre d'applications commerciales.




#### 9.2. Protection des données et des échantillons

Toutes les directives relatives à la protection des données sont rigoureusement respectées. Il est possible que les données doivent être transmises sous forme codée, par exemple pour une publication, et qu'elles puissent être mises à la disposition d'autres chercheur.e.s.

Lorsque des données relatives à la santé ou des échantillons biologiques sont conservés sur place, ils constituent une banque de données ou une biobanque à des fins de recherche. Il se peut que ces données et ces échantillons soient envoyés sous forme codée dans le cadre de ce projet de recherche à une autre banque de données/biobanque. Vous pouvez demander la liste des institutions collaboratrices à la médecin investigatrice/au médecin investigateur.

Le promoteur doit s'assurer que le pays de destination garantit une protection des données équivalente à celle garantie en Suisse.

#### 9.3. Protection des données en cas de réutilisation

Les données et les échantillons de la patiente/du patient pourraient ultérieurement se révéler importants pour répondre à d'autres questionnements et/ou être envoyés à une autre banque de données/biobanque située en Suisse ou à l'étranger pour être aussi exploités dans d'autres projets de recherche (réutilisation). Cette banque de données/biobanque doit toutefois obéir aux mêmes normes et exigences que la banque de données/biobanque du présent projet.

Pour cette réutilisation, en votre qualité de proche ou de représentant e légal e, nous vous prions de signer le document prévu à cet effet (Déclaration de consentement pour la réutilisation de données et échantillons biologiques sous une forme codée). Ce deuxième consentement est indépendant de la participation de la patiente/du patient au projet.

# 9.4. Protection des données en cas d'analyses génétiques

Dès lors que l'on procède à un relevé, un enregistrement ou une transmission de données issues des échantillons de la patiente/du patient dans le cadre de la recherche génétique, il existe des risques liés à la confidentialité (p. ex., la possibilité d'identifier la patiente/le patient), en particulier concernant les informations sur son matériel génétique. Ces risques ne peuvent pas être totalement exclus et augmentent avec la quantité de données pouvant être appariées, notamment si la patiente elle-même/le patient lui-même a publié ou publiera des données génétiques sur Internet (p. ex. à des fins de recherche généalogique). Les informations relatives au matériel génétique de la patiente/du patient peuvent également être importantes pour les membres de sa famille ou sa planification familiale. Le promoteur prend toutes les mesures nécessaires pour réduire le plus possible les risques liés à la confidentialité pour la patiente/le patient.

# 9.5. Droit de consultation dans le cadre d'inspections

Le projet peut faire l'objet d'inspections. Celles-ci peuvent être effectuées par la commission d'éthique compétente ou par le promoteur qui a initié le projet. La médecin-investigatrice/le médecin-investigateur doit alors communiquer les données de la patiente/du patient pour les besoins de ces inspections. Toutes les personnes impliquées sont tenues au plus strict secret professionnel.

## 10. Retrait du projet

La patiente/le patient peut à tout moment se retirer du projet et mettre fin à sa participation si elle/s'il le souhaite ou que vous en décidiez ainsi en tant que proche ou représentant·e légal·e. Les données médicales recueillies jusque-là seront tout de même analysées car une fois intégrées à la base de données leur destruction devient impossible. La patiente/le patient ou vous-même en tant que proche ou représentant·e légal·e pourrez choisir sur la déclaration de retrait de consentement de l'étude @neurIST si :

les données doivent être gardées sous forme codée (codée signifie que le matériel biologique et les données ne peuvent être mis en relation avec la patiente/le patient qu'au moyen d'une clé) ou anonymisée (anonymisée signifie que le code reliant les données à la patiente/au patient sera effacé, plus personne ne pourra savoir que ces données et ces échantillons sont ceux de la patiente/du patient). Ce procédé vise avant tout à assurer la protection de données ;




les échantillons doivent être conservés ou détruits.

#### 11. Rémunération

La patiente/le patient ne percevra aucune rémunération pour sa participation à ce projet de recherche.

Les dépenses telles que les frais de transport qui découlent exclusivement de la participation au projet sont remboursées.

Les prises de sang et les prélèvements de salive et de selles faits uniquement pour ce projet seront prises en charge par @neurIST.

Votre participation n'aura aucune conséquence financière pour vous ou votre assurance maladie. Dans certains cas, les résultats de ce projet peuvent aider à développer des produits commerciaux. Si vous consentez à la participation de la patiente/du patient à ce projet, vous acceptez qu'elle/il renonce dans le même temps à tout droit d'exploitation commerciale (découlant de brevets en particulier).

#### 12. Responsabilité

Les Hôpitaux Universitaire de Genève qui ont initié le projet de recherche et sont chargés de sa réalisation sont responsables des dommages que pourrait subir la patiente/le patient en relation avec le projet. Les conditions et la procédure sont fixées par la loi. Tous les actes étudiés dans cette étude font partie de la pratique quotidienne et relève de standards médicaux ne nécessitant pas une assurance spécifique à l'étude. La responsabilité civile de l'hôpital couvre les dommages éventuels imputables au projet que la patiente/le patient pourrait subir. Si la patiente/le patient subit un dommage du fait de sa participation au projet, il vous faudrait vous adresser au responsable du projet, le Dr Bijlenga.

#### 13. Financement

Le projet est financé par des sources publiques pour l'exploitation académique des données. La coordination du financement est assurée par le bureau @neurIST de la Société européenne pour les traitements neurologiques minimalement invasifs ESMINT (www.esmint.eu). Il est actuellement financé par l'initiation continue de nouveaux projets déposés au Fonds National Suisse pour la recherche ainsi que dans d'autres organismes finançant la recherche en Europe.

#### 14. Interlocuteur(s)

Vous pouvez à tout moment poser des questions au sujet du projet. En cas d'incertitudes pendant ou après le projet, vous pouvez vous adresser à :

Dr Philippe Bijlenga, responsable du projet : 079 204 40 43

Secrétariat du Dr Bijlenga : 022 372 34 26 En écrivant à aneurist : ccc@hcuge.ch

En consultant notre site internet : www.aneurist.org




## Déclaration de consentement

# Déclaration de consentement écrite pour la participation à un projet de recherche

Veuillez lire attentivement ce formulaire. N'hésitez pas à poser des questions lorsque vous ne comprenez pas quelque chose ou que vous souhaitez avoir des précisions. Votre consentement écrit est nécessaire pour la participation de la patiente/du patient au projet.

| Numéro BASEC du projet de recherche (après soumission à la commission d'éthique compétente) : | 2022-00426 |
|---|---|
| Titre<br>(scientifique et usuel) : | @neurIST: informatique biomédicale intégrée pour la gestion des anévrismes cérébraux |
| Institution responsable (responsable du projet et adresse complète) : | Hôpitaux Universitaire de Genève<br>Rue Micheli-du-Crest 24<br>1211 Genève 14 |
| Lieu de réalisation : | Genève, Suisse |
| Responsable du projet sur le site :<br>Nom et prénom en caractères d'imprimerie : | Dr Philippe Bijlenga |
| Participant :<br>Nom et prénom en caractères d'imprimerie :<br>Date de naissance : | |

- En ma qualité de proche ou de représentant·e légal·e de la patiente/du patient susmentionné·e, j'ai obtenu les informations écrites et orales de la part de la médecin-investigatrice/du médecin-investigateur soussigné·e sur les objectifs et le déroulement du projet de recherche ainsi que les avantages et les inconvénients possibles et les risques éventuels.
- Je confirme prendre la décision dans le sens du proche ou de la personne placée sous ma responsabilité, à savoir, qu'elle/qu'il participe au projet de recherche. En son nom, j'accepte les informations écrites et orales. J'ai eu suffisamment de temps pour prendre ma décision.
- J'ai reçu les réponses aux questions que j'ai posées en relation avec la participation à ce projet. Je conserve la feuille d'information et reçois une copie de ma déclaration de consentement.
- J'accepte que les spécialistes compétents de la direction de ce projet et de la commission d'éthique compétente puissent consulter les données non codées de la patiente/du patient afin de procéder à des contrôles et des inspections, à condition toutefois que la confidentialité de ces données soit strictement assurée.
- Je serai informé e en lieu et place de la patiente/du patient des résultats ayant une incidence directe sur sa santé. Si j'estime que cela ne correspond pas à la volonté de la participante/du participant au projet, j'en avise la médecin-investigatrice/le médecin-investigateur du projet.
- Si la patiente/le patient bénéficie / devais bénéficier d'un traitement médical en dehors de l'institution responsable de ce projet, j'accepte que le médecin responsable du projet contacte la/le médecin traitant e de la patiente/du patient et que celui-ci lui fournisse des données médicales concernant la patiente/le patient pouvant être pertinentes pour ce projet.




- Je sais que les données personnelles et les échantillons peuvent être transmis à des fins de recherche dans le cadre de ce projet et uniquement sous une forme codée. Le promoteur assure une protection des données conforme aux normes et exigences Suisses.
- Au nom de la patiente/du patient, je peux, à tout moment et sans avoir à me justifier, révoquer son consentement à la participation, sans que cette décision n'ait de répercussions défavorables sur la suite de sa prise en charge. Les données et les échantillons recueillis jusqu'au retrait seront cependant analysés dans le cadre du projet.
- Je suis informé·e que les HUG sont responsable des dommages éventuels imputables au projet.
- Je suis conscient·e que les obligations mentionnées dans la feuille d'information destinée aux participant·e·s doivent être respectées pendant toute la durée du projet. La médecin-investigatrice/le médecin-investigateur peut exclure la patiente/le patient du projet à tout moment dans l'intérêt de sa santé.

| 0 | Je consens que la patiente/le patient sus-mentionné·e participe à cette étude, j'accepte de donner accès à son dossier de santé, qu'un lien soit créé entre ce dossier et la base de données locale @neurIST, et de remplir un questionnaire sur son histoire clinique : Oui Non |
|---|---|
| 0 | J'accepte que la patiente/le patient sus-mentionné·e fournisse à @neurIST des données sous forme de clichés : ☐ Oui ☐ Non |
| 0 | J'accepte que des échantillons biologiques retirés dans un but thérapeutique à la patiente/le patient sus-mentionné·e soient étudiés : ☐ Oui ☐ Non |
| 0 | J'accepte que la patiente/le patient sus-mentionné·e fournisse des échantillons de sang selon le protocole : ☐ Oui Non |
| 0 | J'accepte que la patiente/le patient sus-mentionné·e fournisse des échantillons de salive selon le protocole : ☐ Oui Non |
| 0 | J'accepte que la patiente/le patient sus-mentionné·e fournisse des échantillons de selles selon le protocole : ☐ Oui Non |
| 0 | J'accepte d'être recontacté·e par @neurIST en vue d'autres consentements ou pour fournir de plus amples informations : Oui Non |




| 0 | médecin traitant·e de la p<br>l'équipe du projet afin d'o | pourrai pas être contacté·e pendant 3 mois, j'accepte que la/le atiente/du patient puisse être contacté·e par un membre de obtenir de sa part des renseignements et des informations statuer sur l'évolution de l'affection cérébro-vasculaire de la |
|---|---|---|
| 0 | Je voudrais que la/le méd participation à cette étude : Oui Non | ecin traitant·e de la patiente/du patient soit informé·e de sa |
| de la r | recherche susceptibles d'être<br>lient ne pas être disponibles a<br>Ces résultats seront mis dan<br>Ces résultats peuvent sig<br>apparentées à la patiente/au<br>La patiente/le patient devra | avant de décider si vous souhaitez être informé·e des résultats pertinents pour la santé de la patiente/du patient (ces résultats avant 4 ans): Ins le dossier médical de la patiente/du patient. Ignaler l'existence d'un risque chez les personnes qui sont u patient, et donc avoir des incidences sur sa famille. Ipeut-être subir de nouveaux tests. Int évoquer des inquiétudes justifiant de recevoir un soutien |
| 0 | Je souhaite être informé·e par la médecin-investigatrice/le médecin-investigateur des résultats susceptibles de concerner la patiente/le patient : Oui Non | |
| 0 | Je souhaite que la/le médrésultats susceptibles de la/ Oui Non | decin traitant·e de la patiente/du patient soit informé·e des<br>le concerner : |
| Médeo | oin Traitant∙e : Nom, Prénom | |
| Si pas | de médecin traitant·e : autre | personne de contact : Nom, Prénom |
| l'entre | tien informatif a eu lieu et l'a | le la/du représentant·e légal·e : Par la présente, j'atteste que dulte incapable de discernement a consenti à participer à cette d'opposition à sa participation. |
| Lieu, | date | Nom et prénom en caractères d'imprimerie |




| | Relation avec la patiente/le patient : |
|---|---|
| | Personne désignée dans les directives anticipées ou dans un mandat pour cause d'inaptitude Curateur/Curatrice Conjoint·e ou son/sa partenaire enregistré·e et fournissant une assistance personnelle régulière Personne faisant ménage commun avec le/la participant·e et fournissant une assistance personnelle régulière Descendant·e et fournissant une assistance personnelle régulière Père/Mère et fournissant une assistance personnelle régulière Frère/Soeur et fournissant une assistance personnelle régulière Signature de la/du proche ou de la/du représentant·e légal·e : |
| avoir expliqué au proche ou à l'importance et la portée du projet projet conformément au droit en réalisation du projet, prendre conformément au droit en réalisation du projet, prendre conformément au droit en réalisation du projet, prendre conformément au droit en réalisation du projet, prendre conformément au droit en reconstruction du projet, prendre conformément au droit en reconstruction du projet en reconstruction du projet et de la portée du projet projet en reconstruction du projet en reconstruction du projet et | stigatrice/du médecin-investigateur : Par la présente, j'atteste la/au représentant·e légal·e du/de la participant·e la nature, . Je déclare satisfaire à toutes les obligations en relation avec ce vigueur. Si je devais, à quelque moment que ce soit durant la naissance d'éléments susceptibles d'influer sur le consentement nt à prendre part au projet, je m'engage à en informer sa/son représentant·e légal·e. |
| Lieu, date | Nom et prénom de la médecin-investigatrice/du médecin-investigateur en caractères d'imprimerie. |
| | Signature de la médecin-investigatrice/du médecin-investigateur : |




Demande de participation à un projet de recherche médical :

## @neurIST: informatique biomédicale intégrée pour la gestion des anévrismes cérébraux

Madame, Monsieur,

La patiente/le patient a été intégré·e à un projet de recherche en situation d'urgence. Selon toute probabilité, elle/il restera durablement incapable de discernement et, par-là, de communiquer sa volonté. Dans la mesure où vous la/le représentez en tant que proche ou représentant·e légal·e, nous vous faisons parvenir le présent document pour vous informer de notre projet de recherche. De plus, nous vous demandons de nous accorder, avec effet rétroactif et en votre qualité de représentant·e, votre consentement pour la participation au projet.

Ci-après, nous vous présentons le projet : d'abord, par un résumé pour vous donner un rapide aperçu ; puis par une description plus détaillée.




Demande de participation à un projet de recherche médical :

# @neurIST : informatique biomédicale intégrée pour la gestion des anévrismes cérébraux

Madame, Monsieur,

Nous vous proposons ici de nous accorder votre consentement pour la participation de la patiente/du patient à notre projet.

La participation est entièrement libre. Toutes les données collectées dans le cadre de ce projet sont soumises à des règles strictes en matière de protection des données.

Le projet de recherche est mené par les Hôpitaux Universitaire de Genève. Nous vous en communiquerons les résultats si vous le souhaitez.

Lors d'un entretien, nous vous présenterons les éléments essentiels et répondrons à vos questions. Pour vous proposer d'ores et déjà un aperçu du projet, voici les points clés à retenir. Vous trouverez à la suite des informations complémentaires plus détaillées.

# Pourquoi menons-nous ce projet de recherche?

- Notre projet porte sur les anévrismes cérébraux qui sont des anomalies observées sur les vaisseaux sanguins irriguant notre cerveau. Les anévrismes cérébraux sont diagnostiqués par radiographie, scanners, angiographie ou IRM. Lors de la rupture d'un anévrisme cérébral, le traitement de cet anévrisme est indispensable pour permettre la survie de la patiente/du patient.
- Notre projet de recherche vise à déterminer les causes et les évolutions des anévrismes cérébraux afin d'améliorer leur prise en charge.

# Que doit faire le patient en cas de participation ? – Que se passe-t-il pour le patient en cas de participation ?

- Forme de la participation : Si vous nous accordez votre consentement pour la participation de la patiente/du patient, nous récolterons des informations générales concernant la patiente/le patient et nous lui prélèverons du sang, de la salive et des selles. Nous conserverons pour la recherche les tissus et le liquide enlevés dans le cadre du traitement de l'anévrisme.
- Déroulement pour les participant·e·s: Si le patient participe au projet, sa participation à cette étude implique, en plus de son suivi habituel, une ou plusieurs prise(s) de sang, le prélèvement de salive et de selles, et un questionnaire sur sa qualité de vie qu'elle/il devra remplir lors de visites de routine. Des informations la/le concernant et concernant son anévrisme seront relevées à partir de son dossier hospitalier. La patiente/le patient pourra aussi être contacté pour fournir des informations complémentaires ou pour donner son autorisation pour d'autres études cliniques.



# Quels sont les bénéfices et les risques liés à la participation au projet ?

# Bénéfices pour les participants

- La participation à ce projet de recherche n'apportera à la patiente/au patient aucun bénéfice direct.
- Par sa participation, la patiente/le patient contribue à aider les futurs patient e.s.

# Risques et contraintes

 Les risques associés à cette étude sont ceux liés à la réalisation d'une prise de sang (risque infectieux faible, hématome) et à l'utilisation d'un réseau informatique pour le transfert des données dont la sécurité ne peut jamais être totalement garantie.

En apposant votre signature à la fin du document, vous attestez en avoir compris tout le contenu et accorder librement votre consentement pour la participation de la patiente/du patient au projet.




### Information détaillée

# 1. Objectif du projet et sélection des participant·e·s

Dans cette feuille d'information, notre projet de recherche est aussi simplement désigné par le terme *projet*. Si vous accordez votre consentement, en votre qualité de proche ou de représentant e légal e, pour la participation du patient, ce dernier est un e participant e au projet.

Ce projet permettra de mieux comprendre les causes et les évolutions des anévrismes cérébraux afin d'améliorer leur prise en charge. Ce projet conduira en effet à la création d'un système informatisé d'aide à la décision pour le traitement des anévrismes cérébraux.

Nous vous sollicitons en votre qualité de proche ou de représentant e légale, car la participation est ouverte à toutes les personnes chez qui un anévrisme cérébral a été diagnostiqué.

# 2. Informations générales sur le projet

Ce projet international regroupant plusieurs centres hospitaliers a débuté en 2006. Les études menées sur les anévrismes cérébraux suggèrent que plusieurs facteurs sont impliqués dans l'apparition et l'évolution de cette maladie. Parmi ces facteurs, nos gènes, nos protéines et notre microbiote (bactéries vivant dans notre bouche et notre système digestif) semblent jouer un rôle important. Bien qu'il ait été montré que des modifications du microbiote par l'alimentation ou la consommation d'antibiotiques influence l'évolution de diverses maladies, son rôle dans l'apparition et l'évolution des anévrismes cérébraux n'est pas clairement défini.

Nous récolterons des informations générales concernant tous les participant·e·s et nous prélèverons du sang, de la salive et des selles.

Nous récolterons également des informations concernant l'anévrisme de la patiente/du patient. Lors de l'intervention pour le traitement de l'anévrisme, une partie de celui-ci a été prélevé, ainsi que du liquide céphalo-rachidien (liquide dans lequel baigne le cerveau). Ces prélèvements ont été effectués dans le cadre de la prise en charge standard et non pas spécifiquement pour le projet. Lors de l'intervention pour le traitement de l'anévrisme, du sang, de la salive et des selles ont été prélevés spécifiquement pour le projet.

Avec votre accord, ces prélèvements seront conservés et utilisés pour le projet.

Ces informations et prélèvements nous permettrons de chercher des facteurs communs susceptibles d'expliquer pourquoi certaines personnes sont plus à risque vis-à-vis des anévrismes que d'autres.

Le nombre de personnes recrutées au HUG pour ce projet sera d'environ 150 patient·e·s par an, 45 membres de la famille par an et 105 volontaires sain·e·s par an. A l'heure actuelle, il est prévu de conserver les informations et les échantillons pour une période initiale de 20 ans.

Ce projet est réalisé dans le respect des prescriptions de la législation Suisse. Nous suivons en outre l'ensemble des directives reconnues au niveau international. La commission d'éthique compétente a examiné et autorisé ce projet.

# 3. Déroulement pour les participant·e·s

- Des informations concernant la patiente/le patient et concernant son anévrisme (scanners, IRM, radiographies et angiogrammes) seront relevées à partir de son dossier hospitalier.
- Des échantillons de sang seront prélevés. La prise de sang sera faite lors d'une visite de routine. Les échantillons de sang seront prélevés soit pour : A) l'étude génétique et l'analyse des modifications d'expression des gènes et des protéines dans le sang (3 échantillons de sang pour un volume maximal de 39 ml), soit B) pour l'étude bactériologique (3 échantillons de sang pour un volume maximal de 17 ml). Lors du traitement de l'anévrisme, une prise de sang a été faite. Une autre pourra être faite dans les 48 heures suivant le traitement de l'anévrisme et lors d'une visite de routine (2 échantillons de sang pour un volume maximal de 22 ml pour




l'analyse des modifications d'expression des gènes et des protéines dans le sang, ou, 3 échantillons de sang pour un volume maximal de 17 ml pour l'analyse bactériologique).

- Un échantillon de salive a été prélevé lors du traitement de l'anévrisme. Un autre échantillon sera prélevé lors d'une visite de routine après le traitement de l'anévrisme (6 mois après l'arrêt de tout traitement antibiotique).
- Un échantillon de selles a été prélevé lors du traitement de l'anévrisme. Un autre échantillon sera prélevé lors d'une visite de routine après le traitement de l'anévrisme (6 mois après l'arrêt de tout traitement antibiotique).
- Lors du traitement de l'anévrisme de la patiente/du patient, une partie de celui-ci a été prélevé, ainsi que du liquide céphalo-rachidien. Ces prélèvements sont effectués dans le cadre de la prise en charge standard et non pas spécifiquement pour le projet. Avec votre accord, ces prélèvements seront conservés pour le projet.
- Il sera demandé à la patiente/au patient de compléter, avec assistance (pour s'assurer de la compréhension), un questionnaire sur sa qualité de vie (durée d'environ 30 minutes). Ce questionnaire lui sera donné lors de sa première visite et lors des visites de routine effectuées pour le contrôle de son anévrisme.
- Vous pourrez aussi être contacté·e en dehors des visites de routine de la patiente/du patient, soit pour vous demander des informations complémentaires, soit pour vous proposer que la patiente/le patient participe à d'autres études cliniques.

Il se peut que nous devions retirer la patiente/le patient du projet avant le terme prévu. Cette situation peut se produire si le projet est interrompu précocement et qu'il est demandé que les données soient détruites.

Avec votre accord, la médecin traitante/le médecin traitant sera informé de la participation de la patiente/du patient à ce projet.

## 4. Bénéfices pour les participant·e·s

La participation à ce projet de recherche n'apportera pas de bénéfice personnel à la patiente/au patient.

Les résultats des recherches pourraient se révéler importants par la suite pour les personnes touchées par la même maladie.

#### 5. Caractère facultatif de la participation et obligations

La participation au projet de recherche est entièrement libre. Si la patiente/le patient ne souhaite pas participer ou si vous, en tant que proche ou représentant·e légal·e, revenez ultérieurement sur votre décision à ce sujet, vous n'aurez pas à vous justifier. Cette décision n'aura pas de répercussions défavorables sur la suite de sa prise en charge médicale.

La participation au projet implique les obligations suivantes :

- la patiente/le patient est tenu·e de suivre les instructions et de remplir les exigences prévues par le protocole de recherche ;
- la médecin investigatrice/le médecin-investigateur doit être informé·e de l'évolution de la maladie et il convient de lui signaler tout nouveau symptôme, tout nouveau trouble et tout changement dans l'état de la patiente/du patient :
- la médecin investigatrice/le médecin-investigateur doit être informé·e de tout traitement ou thérapie prescrit par un·e autre médecin ainsi que de tous les médicaments pris par la patiente/le patient, même sans ordonnance.

#### 6. Risques et contraintes pour les participantes

En participant au projet, la patiente/le patient ne sera exposé·e qu'à des risques mineurs tels qu'une prise de sang (risque infectieux faible, hématome) et à l'utilisation d'un réseau informatique pour le transfert des données dont la sécurité ne peut jamais être totalement garantie.

Nous nous efforcerons de rendre les prises de sang aussi peu douloureuses que possible et mettrons en place des mesures de sécurité pour tous nos transferts de données codées.




Si certains résultats issus du projet (découverte de maladies lors des examens radiologiques ou sanguins) étaient susceptibles d'engendrer des inquiétudes chez la patiente/le patient, nous lui proposerons un soutien psychologique.

#### 7. Alternatives

Si vous ne souhaitez pas que la patiente/le patient participe à ce projet de recherche, mais vous restez ouvert à la possibilité d'une participation à d'autres projets, merci de l'indiquer informer la médecin-investigatrice/le médecin-investigateur.

#### 8. Résultats

Le projet permet d'obtenir différents résultats :

- 1. des résultats individuels qui concernent directement la patiente/le patient,
- 2. des résultats individuels découverts par hasard (ce qu'on appelle les découvertes fortuites),
- 3. les résultats définitifs objectifs du projet dans son ensemble.
- 1. Au cours du projet, la médecin-investigatrice/le médecin-investigateur vous avisera, en votre qualité de proche ou de représentant·e légal·e, de toute nouvelle découverte importante pour la patiente/le patient. Vous serez informé·e oralement et par écrit ; vous pourrez par la suite à nouveau décider si la patiente/le patient doit poursuivre sa participation au projet.
- 2. Les découvertes fortuites constituent des « résultats concomitants », à savoir des résultats qui n'ont pas été explicitement recherchés, mais qui ont été obtenus par hasard. Il peut s'agir p. ex. de résultats d'analyses génétiques ou de procédés d'imagerie.

Vous serez informé·e des découvertes fortuites si elles ont une incidence sur la santé de la patiente/du patient. Cela signifie que ces découvertes sont communiquées si l'on constate par hasard une pathologie qui n'était pas encore connue jusqu'alors ou que l'on peut empêcher l'apparition d'une maladie par des mesures de prévention. Si vous ne souhaitez pas recevoir ces informations (« droit de ne pas savoir »), merci de l'indiquer à la médecin-investigatrice/au médecin-investigateur.

Certains résultats pourraient nécessiter un test de confirmation. Une fois confirmés, ces résultats seront directement ajoutés au dossier médical de la patiente/du patient et pourraient donc être consultés par toute personne à qui la patiente/le patient a donné accès au dossier (par exemple, un employeur ou une compagnie d'assurance).

3. La médecin-investigatrice/le médecin-investigateur peut vous faire parvenir, à l'issue du projet, une synthèse des résultats globaux.

#### 9. Confidentialité des données et des échantillons

#### 9.1. Traitement et codage des données

Dans le cadre de ce projet de recherche, des données relatives à la santé de la patiente/du patient sont recueillies et traitées, en partie de manière automatisée. Ces informations sont codées au moment du relevé. Le codage signifie que toutes les données permettant d'identifier la patiente/le patient (nom, date de naissance, etc.) sont effacées et remplacées par un code. Il n'est pas possible de relier les données à la patiente/au patient sans le code, qui reste en permanence au sein des Hôpitaux Universitaire de Genève.

Seul un nombre limité de personnes peut consulter les données de la patiente/du patient sous une forme non codée, et ce, exclusivement pour pouvoir accomplir les tâches nécessaires au déroulement du projet de recherche. Ces personnes sont tenues au secret professionnel. En votre qualité de proche ou représentant e légal e, vous avez le droit de consulter les données de la patiente/du patient.

La base de données proprement dite sera également conservée après la fin de @neurIST et pourra être mise à disposition, sous forme codée, à d'autres chercheurs, éventuellement contre rémunération, voire développée dans le cadre d'applications commerciales.




#### 9.2. Protection des données et des échantillons

Toutes les directives relatives à la protection des données sont rigoureusement respectées. Il est possible que les données doivent être transmises sous forme codée, par exemple pour une publication, et qu'elles puissent être mises à la disposition d'autres chercheur.e.s.

Lorsque des données relatives à la santé ou des échantillons biologiques sont conservés sur place, ils constituent une banque de données ou une biobanque à des fins de recherche. Il se peut que ces données et ces échantillons soient envoyés sous forme codée dans le cadre de ce projet de recherche à une autre banque de données/biobanque. Vous pouvez demander la liste des institutions collaboratrices à la médecin investigatrice/au médecin investigateur.

Le promoteur doit s'assurer que le pays de destination garantit une protection des données équivalente à celle garantie en Suisse.

# 9.3. Protection des données en cas de réutilisation

Les données et les échantillons de la patiente/du patient pourraient ultérieurement se révéler importants pour répondre à d'autres questionnements et/ou être envoyés à une autre banque de données/biobanque située en Suisse ou à l'étranger pour être aussi exploités dans d'autres projets de recherche (réutilisation). Cette banque de données/biobanque doit toutefois obéir aux mêmes normes et exigences que la banque de données/biobanque du présent projet.

Pour cette réutilisation, en votre qualité de proche ou de représentant e légal e, nous vous prions de signer le document prévu à cet effet (Déclaration de consentement pour la réutilisation de données et échantillons biologiques sous une forme codée). Ce deuxième consentement est indépendant de la participation de la patiente/du patient au projet.

# 9.4. Protection des données en cas d'analyses génétiques

Dès lors que l'on procède à un relevé, un enregistrement ou une transmission de données issues des échantillons de la patiente/du patient dans le cadre de la recherche génétique, il existe des risques liés à la confidentialité (p. ex., la possibilité d'identifier la patiente/le patient), en particulier concernant les informations sur son matériel génétique. Ces risques ne peuvent pas être totalement exclus et augmentent avec la quantité de données pouvant être appariées, notamment si la patiente elle-même/le patient lui-même a publié ou publiera des données génétiques sur Internet (p. ex. à des fins de recherche généalogique). Les informations relatives au matériel génétique de la patiente/du patient peuvent également être importantes pour les membres de sa famille ou sa planification familiale. Le promoteur prend toutes les mesures nécessaires pour réduire le plus possible les risques liés à la confidentialité pour la patiente/le patient.

# 9.5. Droit de consultation dans le cadre d'inspections

Le projet peut faire l'objet d'inspections. Celles-ci peuvent être effectuées par la commission d'éthique compétente ou par le promoteur qui a initié le projet. La médecin-investigatrice/le médecin-investigateur doit alors communiquer les données de la patiente/du patient pour les besoins de ces inspections. Toutes les personnes impliquées sont tenues au plus strict secret professionnel.

# 10. Retrait du projet

La patiente/le patient peut à tout moment se retirer du projet et mettre fin à sa participation si elle/s'il le souhaite ou que vous en décidiez ainsi en tant que proche ou représentant·e légal·e. Les données médicales recueillies jusque-là seront tout de même analysées car une fois intégrées à la base de données leur destruction devient impossible. La patiente/le patient ou vous-même en tant que proche ou représentant·e légal·e pourrez choisir sur la déclaration de retrait de consentement de l'étude @neurIST si :

o les données doivent être gardées sous forme codée (codée signifie que le matériel biologique et les données ne peuvent être mis en relation avec la patiente/le patient qu'au moyen d'une clé) ou anonymisée (anonymisée signifie que le code reliant les données à la patiente/au patient sera effacé, plus personne ne pourra savoir que ces données et ces




échantillons sont ceux de la patiente/du patient). Ce procédé vise avant tout à assurer la protection de données ;

o les échantillons doivent être conservés ou détruits.

#### 11. Rémunération

La patiente/le patient ne percevra aucune rémunération pour sa participation à ce projet de recherche.

Les dépenses telles que les frais de transport qui découlent exclusivement de la participation au projet sont remboursées.

Les prises de sang et les prélèvements de salive et de selles faits uniquement pour ce projet seront prises en charge par @neurIST.

Votre participation n'aura aucune conséquence financière pour vous ou votre assurance maladie. Dans certains cas, les résultats de ce projet peuvent aider à développer des produits commerciaux. Si vous consentez à la participation de la patiente/du patient à ce projet, vous acceptez qu'elle/il renonce dans le même temps à tout droit d'exploitation commerciale (découlant de brevets en particulier).

## 12. Responsabilité

Les Hôpitaux Universitaire de Genève qui ont initié le projet de recherche et sont chargés de sa réalisation sont responsables des dommages que pourrait subir la patiente/le patient en relation avec le projet. Les conditions et la procédure sont fixées par la loi. Tous les actes étudiés dans cette étude font partie de la pratique quotidienne et relève de standards médicaux ne nécessitant pas une assurance spécifique à l'étude. La responsabilité civile de l'hôpital couvre les dommages éventuels imputables au projet que la patiente/le patient pourrait subir. Si la patiente/le patient subit un dommage du fait de sa participation au projet, il vous faudrait vous adresser au responsable du projet, le Dr Bijlenga.

### 13. Financement

Le projet est financé par des sources publiques pour l'exploitation académique des données. La coordination du financement est assurée par le bureau @neurIST de la Société européenne pour les traitements neurologiques minimalement invasifs ESMINT (www.esmint.eu). Il est actuellement financé par l'initiation continue de nouveaux projets déposés au Fonds National Suisse pour la recherche ainsi que dans d'autres organismes financant la recherche en Europe.

# 14. Interlocuteur(s)

Vous pouvez à tout moment poser des questions au sujet du projet. En cas d'incertitudes pendant ou après le projet, vous pouvez vous adresser à :

Dr Philippe Bijlenga, responsable du projet : 079 204 40 43

Secrétariat du Dr Bijlenga : 022 372 34 26 En écrivant à aneurist : ccc@hcuge.ch

En consultant notre site internet : www.aneurist.org




### Déclaration de consentement

## Déclaration de consentement écrite pour la participation à un projet de recherche

Veuillez lire attentivement ce formulaire. N'hésitez pas à poser des questions lorsque vous ne comprenez pas quelque chose ou que vous souhaitez avoir des précisions. Votre consentement écrit est nécessaire pour la participation de la patiente/du patient au projet.

| Numéro BASEC du projet de recherche (après soumission à la commission d'éthique compétente) : | 2022-00426 |
|---|---|
| Titre<br>(scientifique et usuel) : | @neurIST: informatique biomédicale intégrée pour la gestion des anévrismes cérébraux |
| Institution responsable (responsable du projet et adresse complète) : | Hôpitaux Universitaire de Genève<br>Rue Micheli-du-Crest 24<br>1211 Genève 14 |
| Lieu de réalisation : | Genève, Suisse |
| Responsable du projet sur le site :<br>Nom et prénom en caractères d'imprimerie : | Dr Philippe Bijlenga |
| Participant :<br>Nom et prénom en caractères d'imprimerie :<br>Date de naissance : | |

- En ma qualité de proche ou de représentant·e légal·e de la patiente/du patient susmentionné·e, j'ai obtenu les informations écrites et orales de la part de la médecin-investigatrice/du médecin-investigateur soussigné·e sur les objectifs et le déroulement du projet de recherche ainsi que les avantages et les inconvénients possibles et les risques éventuels.
- Je confirme prendre la décision dans le sens du proche ou de la personne placée sous ma responsabilité, à savoir, qu'elle/qu'il participe au projet de recherche. En son nom, j'accepte les informations écrites et orales. J'ai eu suffisamment de temps pour prendre ma décision.
- J'ai reçu les réponses aux questions que j'ai posées en relation avec la participation à ce projet. Je conserve la feuille d'information et reçois une copie de ma déclaration de consentement.
- J'accepte que les spécialistes compétents de la direction de ce projet et de la commission d'éthique compétente puissent consulter les données non codées de la patiente/du patient afin de procéder à des contrôles et des inspections, à condition toutefois que la confidentialité de ces données soit strictement assurée.
- Je serai informé e en lieu et place de la patiente/du patient des résultats ayant une incidence directe sur sa santé. Si j'estime que cela ne correspond pas à la volonté de la participante/du participant au projet, j'en avise la médecin-investigatrice/le médecin-investigateur du projet.
- Si la patiente/le patient bénéficie / devais bénéficier d'un traitement médical en dehors de l'institution responsable de ce projet, j'accepte que le médecin responsable du projet contacte la/le médecin traitant e de la patiente/du patient et que celui-ci lui fournisse des données médicales concernant la patiente/le patient pouvant être pertinentes pour ce projet.




- Je sais que les données personnelles et les échantillons peuvent être transmis à des fins de recherche dans le cadre de ce projet et uniquement sous une forme codée. Le promoteur assure une protection des données conforme aux normes et exigences Suisses.
- Au nom de la patiente/du patient, je peux, à tout moment et sans avoir à me justifier, révoquer son consentement à la participation, sans que cette décision n'ait de répercussions défavorables sur la suite de sa prise en charge. Les données et les échantillons recueillis jusqu'au retrait seront cependant analysés dans le cadre du projet.
- Je suis informé·e que les HUG sont responsable des dommages éventuels imputables au projet.
- Je suis conscient·e que les obligations mentionnées dans la feuille d'information destinée aux participant·e·s doivent être respectées pendant toute la durée du projet. La médecin-investigatrice/le médecin-investigateur peut exclure la patiente/le patient du projet à tout moment dans l'intérêt de sa santé.

| 0 | Je consens que la patiente/le patient sus-mentionné·e participe à cette étude, j'accepte de donner accès à son dossier de santé, qu'un lien soit créé entre ce dossier et la base de données locale @neurIST, et de remplir un questionnaire sur son histoire clinique : Oui Non |
|---|---|
| 0 | J'accepte que la patiente/le patient sus-mentionné·e fournisse à @neurIST des données sous forme de clichés : ☐ Oui ☐ Non |
| 0 | J'accepte que des échantillons biologiques retirés dans un but thérapeutique à la patiente/le patient sus-mentionné·e soient étudiés : ☐ Oui ☐ Non |
| 0 | J'accepte que la patiente/le patient sus-mentionné·e fournisse des échantillons de sang selon le protocole : ☐ Oui Non |
| 0 | J'accepte que la patiente/le patient sus-mentionné·e fournisse des échantillons de salive selon le protocole : ☐ Oui Non |
| 0 | J'accepte que la patiente/le patient sus-mentionné·e fournisse des échantillons de selles selon le protocole : ☐ Oui ☐ Non |
| 0 | J'accepte d'être recontacté·e par @neurIST en vue d'autres consentements ou pour fournir de plus amples informations : Oui Non |




| 0 | Dans l'hypothèse où je ne pourrai pas être contacté·e pendant 3 mois, j'accepte que la/le médecin traitant·e de la patiente/du patient puisse être contacté·e par un membre de l'équipe du projet afin d'obtenir de sa part des renseignements et des informations médicales permettant de statuer sur l'évolution de l'affection cérébro-vasculaire de la patiente/du patient : Oui Non |
|---|---|
| 0 | Je voudrais que la/le médecin traitant·e de la patiente/du patient soit informé·e de sa participation à cette étude : Oui Non |
| de la r | ez étudier les points suivants avant de décider si vous souhaitez être informé·e des résultats echerche susceptibles d'être pertinents pour la santé de la patiente/du patient (ces résultats ient ne pas être disponibles avant 4 ans): Ces résultats seront mis dans le dossier médical de la patiente/du patient. Ces résultats peuvent signaler l'existence d'un risque chez les personnes qui son apparentées à la patiente/au patient, et donc avoir des incidences sur sa famille. La patiente/le patient devra peut-être subir de nouveaux tests. Certains résultats pourraient évoquer des inquiétudes justifiant de recevoir un soutier psychologique. |
| 0 | Je souhaite être informé·e par la médecin-investigatrice/le médecin-investigateur des résultats susceptibles de concerner la patiente/le patient: Oui Non |
| 0 | Je souhaite que la/le médecin traitant·e de la patiente/du patient soit informé·e des résultats susceptibles de la/le concerner : Oui Non |
| Médeo | sin Traitant·e : Nom, Prénom |
| Si pas | de médecin traitant·e : autre personne de contact : Nom, Prénom |
| l'entre | ation de la/du proche ou de la/du représentant·e légal·e : Par la présente, j'atteste que tien informatif a eu lieu et l'adulte incapable de discernement a consenti à participer à cette et/ou qu'il n'y a aucun signe d'opposition à sa participation. |
| Lieu, | Nom et prénom en caractères d'imprimerie |




| | Relation avec la patiente/le patient : |
|---|---|
| | Personne désignée dans les directives anticipées ou dans un mandat pour cause d'inaptitude Curateur/Curatrice Conjoint·e ou son/sa partenaire enregistré·e et fournissant une assistance personnelle régulière Personne faisant ménage commun avec le/la participant·e et fournissant une assistance personnelle régulière Descendant·e et fournissant une assistance personnelle régulière Père/Mère et fournissant une assistance personnelle régulière Frère/Soeur et fournissant une assistance personnelle régulière Signature de la/du proche ou de la/du représentant·e légal·e : |
| avoir expliqué au proche ou à<br>l'importance et la portée du projet.<br>projet conformément au droit en<br>éalisation du projet, prendre conr | tigatrice / du médecin-investigateur : Par la présente, j'atteste la/au représentant·e légal·e du/de la participant·e la nature, Je déclare satisfaire à toutes les obligations en relation avec ce vigueur. Si je devais, à quelque moment que ce soit durant la naissance d'éléments susceptibles d'influer sur le consentement t à prendre part au projet, je m'engage à en informer sa/son représentant·e légal·e. |
| | Nom et prénom de la médecin-investigatrice/du médecin-investigateur en caractères d'imprimerie. |
| | Signature de la médecin-investigatrice/du médecin-investigateur : |




# Confirmation écrite d'un médecin non associé au projet de recherche

Confirmation écrite pour le médecin non associé au projet de recherche, qui *n'*est *pas* impliqué dans le projet de recherche mentionné ci-après et qui défend les intérêts de la personne se prêtant à l'expérience (LRH art 30).

# Données sur le projet de recherche

| Titre du projet de recherche: @neurIST : informatique biomédicale intégrée pour la gestion des anévrismes cérébraux | |
|---|---|
| Numéro du projet de recherche: | |
| Lieu où se déroule le projet de recherche : Hôpit | aux Universitaire de Genève |
| Nom et prénom du médecin investigateur respor | nsable: Bijlenga Philippe |
| Nom et prénom du / de la participant·e: | |
| Date de naissance (facultatif): | sexe (facultatif): |

J'ai reçu et j'ai lu le résumé du protocole du projet de recherche susmentionné.

J'atteste que les intérêts du / de la participant e sont respectés et que son suivi médical est garanti.

| Lieu, date | Nom, prénom et numéro de téléphone<br>du médecin non associé au projet de<br>recherche (en caractères d'imprimerie) | Signature du médecin non associé au projet de recherche |
|---|---|---|

Par la présente, j'atteste avoir expliqué au médecin non associé au projet de recherche la nature, l'importance et la portée du projet. Si je devrai prendre connaissance, à quelque moment que ce soit durant la réalisation du projet, d'éléments susceptibles d'influer sur le consentement du / de la participant e à prendre part au projet de recherche, je m'engage à l'en informer immédiatement.

| Lieu, date | Nom, prénom et numéro de téléphone<br>de l'investigateur responsable (en<br>caractères d'imprimerie) | Signature de l'investigateur responsable |
|---|---|---|
|---|---|---|




@neurIST : informatique biomédicale intégrée pour la gestion des anévrismes cérébraux Ce projet est organisé par : Hôpitaux Universitaire Genève

Madame, Monsieur,

Nous vous proposons de participer à notre projet de recherche.

La présente notice d'information est destinée à être lue en parallèle avec la notice générale d'information destinée aux participant·e·s, qui doit également vous avoir été remise. Cette feuille d'information ne décrit que les points spécifiques aux tests génétiques.

### 1. Objectifs de l'étude génétique

Des résultats préliminaires publiés dans la littérature montrent que des facteurs génétiques, en parallèle des facteurs environnementaux, pourraient contribuer à l'apparition et au développement des anévrismes, cependant leurs rôles précis ne sont pas encore élucidés. Le but des tests génétiques au sein de notre étude @neurIST est donc d'identifier les gènes qui seraient impliqués dans les anévrismes cérébraux.

## 2. Déroulement pour les participants

Une analyse génétique couvrant tout votre génome sera effectuée sur votre échantillon sanguin prélevé lors d'une consultation avec votre clinicien ou avec la médecin-investigatrice/le médecin-investigateur.

Les gènes des patient·e·s présentant des anévrismes cérébraux seront comparés aux gènes de sujets contrôles (participant·e inclus·e dans l'étude en tant que « Membre de la famille » ou en tant que « Volontaire sain·e ») afin de découvrir des variantes dans le génome des patients qui pourraient être associées à une susceptibilité plus importante pour les anévrismes cérébraux.

Si vous faites partie de l'étude familiale, l'ensemble de votre génome sera comparé à celui d'autres membres de votre famille afin également de découvrir des gènes candidats liés aux anévrismes.

Ces gènes candidats seront ensuite utilisés pour tester les échantillons de sang remis par des patient·e·s présentant un anévrisme. Les résultats de ces expériences seront placés dans des bases de données informatisées sécurisées. Leur analyse pourrait prendre jusqu'à dix ans.

#### 3. Risques

Les risques associés à cette étude sont ceux liés à la réalisation d'une prise de sang (risque infectieux faible, hématome) et l'utilisation d'un réseau informatique pour le transfert des données dont la sécurité ne peut jamais être totalement garantie.

Nous nous efforcerons de rendre les prises de sang aussi peu douloureuses que possible et mettrons en place des mesures de sécurité pour tous nos transferts de données codées.

Un risque associé à l'étude génétique est la découverte fortuite d'une anomalie associée à une maladie connue. Si certains résultats issus de cette étude génétique étaient susceptibles d'engendrer des inquiétudes chez vous, nous vous proposerons un soutien psychologique.

#### 4. Découvertes pendant l'étude génétique

Toute découverte survenant durant l'étude et pertinente pour votre santé vous sera communiquée. Si vous ne souhaitez pas obtenir ce type d'information, veuillez en aviser la médecin-investigatrice/le médecin-investigateur.

Ces résultats génétiques peuvent avoir un impact sur votre famille, avec laquelle vous partagez certains gènes. Si ce cas de figure survient, nous discuterons avec vous sur comment informer les autres membres de la famille.

Si vous participez à l'étude familiale, les tests pourraient également révéler des cas de non-paternité ; ces résultats ne seront communiqués ni à vous-même ni aux autres membres de votre famille.

Version du 12.07.2022



### 5. Confidentialité des données et des échantillons biologiques

D'une manière générale, le traitement et codages des données, ainsi que la protection des données et des échantillons sont similaires à ce qui est décrit dans la lettre d'information générale qui vous a été donnée dans le cadre du projet @neurIST.

Concernant le cas particulier de la protection des données en cas d'analyses génétiques : Dès lors que l'on procède à un relevé, un enregistrement ou une transmission de données issues de vos échantillons dans le cadre de la recherche génétique, il existe des risques liés à la confidentialité (p. ex., la possibilité de vous identifier), en particulier concernant les informations sur votre matériel génétique. Ces risques ne peuvent pas être totalement exclus et augmentent avec la quantité de données pouvant être appariées, notamment si vous publiez vous-même des données génétiques sur Internet (p. ex. à des fins de recherche généalogique). Les informations relatives à votre matériel génétique peuvent également être importantes pour les membres de votre famille ou votre planification familiale. Le promoteur prend toutes les mesures nécessaires pour réduire le plus possible les risques liés à la confidentialité.

# 6. Participation à l'étude génétique et retrait de l'étude

Vous pouvez décider de ne pas participer à l'étude génétique @neurIST, tout en fournissant d'autres informations à l'étude. Si vous décidez de ne pas participer, cela ne changera rien à votre prise en charge médicale, de votre anévrisme le cas échéant. Vous n'avez pas à justifier vos décisions.

Vous pouvez à tout moment vous retirer de l'étude génétique si vous le souhaitez. Vous n'avez pas à justifier vos décisions. Les données médicales recueillies jusque-là seront tout de même analysées car une fois intégrées à la base de données leur destruction devient impossible. Vous pourrez choisir si vous souhaitez que :

- vos données soient gardées sous forme codée (codée signifie que mon matériel biologique et mes données ne peuvent être mis en relation avec ma personne qu'au moyen d'une clé) ou anonymisée (anonymisée signifie que le code reliant mes données à ma personne sera effacé, plus personne ne pourra savoir que ces données et ces échantillons sont les miens)
- vos échantillons biologiques soient conservés ou détruits.

# 7. Interlocuteurs

Vous pouvez à tout moment poser vos questions et demander toutes les précisions nécessaires en vous adressant au :

Dr Philippe Bijlenga, responsable du projet : 079 204 40 43

Secrétariat du Dr Bijlenga : 022 372 34 26 En écrivant à aneurist : ccc@hcuge.ch

En consultant notre site internet : www.aneurist.org



# Déclaration de consentement pour l'étude génétique @neurIST

Veuillez lire attentivement ce formulaire. N'hésitez pas à poser des questions lorsque vous ne comprenez pas quelque chose ou que vous souhaitez avoir des précisions. Votre consentement écrit est nécessaire pour participer au projet.

| Numéro BASEC du projet :<br>(après soumission à la commission d'éthique<br>compétente) : | 2022-00426 |
|---|---|
| Titre de l'étude :<br>(titre scientifique et titre usuel) | @neurIST : informatique biomédicale intégrée pour la gestion des anévrismes cérébraux |
| Institution responsable : (adresse complète) : | Hôpitaux Universitaire de Genève<br>Rue Micheli-du-Crest 24<br>1211 Genève 14 |
| Lieu de réalisation du projet : | Genève, Suisse |
| Directeur du projet sur le site :<br>(nom et prénom en caractères d'imprimerie) : | Dr Philippe Bijlenga |
| Participant / participante :<br>(nom et prénom en caractères d'imprimerie) :<br>Date de naissance : | |

- Je déclare avoir été informé·e, par la médecin-investigatrice/le médecin-investigateur soussigné·e, oralement et par écrit, des objectifs et du déroulement du projet ainsi que des effets présumés, des avantages, des inconvénients possibles et des risques éventuels.
- Je prends part à ce projet de façon volontaire et j'accepte le contenu de la feuille d'information qui m'a été remise sur le projet précité. J'ai eu suffisamment de temps pour prendre ma décision.
- J'ai reçu les réponses aux questions que j'ai posées en relation avec la participation à ce projet. Je conserve la feuille d'information et reçois une copie de ma déclaration de consentement écrite.
- J'accepte que les spécialistes compétent·e·s de la direction de ce projet et de la commission d'éthique compétente puissent consulter mes données non codées afin de procéder à des contrôles et des inspections, à condition toutefois que la confidentialité de ces données soit strictement assurée.
- Si je bénéficie / devais bénéficier d'un traitement médical en dehors de l'institution responsable de ce projet, j'accepte que le médecin responsable du projet contacte ma/mon médecin traitant·e et que celui-ci lui fournisse des données médicales me concernant pouvant être pertinentes pour ce projet.
- Je sais que mes données personnelles, mes données de santé, et mes échantillons peuvent être transmis à des fins de recherche dans le cadre de ce projet et uniquement sous une forme codée. Le promoteur assure une protection des données conforme aux normes et exigences Suisses.
- Je peux, à tout moment et sans avoir à me justifier, révoquer mon consentement à participer au projet, sans que cette décision n'ait de répercussions défavorables sur la suite de ma prise en charge. Les données et les échantillons recueillis jusqu'au retrait seront cependant analysés dans le cadre du projet.
- Je suis informé·e que les Hôpitaux Universitaire Genevois sont responsables des dommages éventuels imputables au projet.
- Je suis conscient·e que les obligations mentionnées dans la feuille d'information destinée aux participant·e·s doivent être respectées pendant toute la durée du projet. La médecin-



investigatrice/le médecin-investigateur peut m'exclure à tout moment du projet dans l'intérêt de ma santé.

Je consens à participer à cette étude.

Veuillez étudier les points suivants avant de décider si vous souhaitez être informé des résultats de la recherche susceptibles d'être pertinents pour votre santé (ces résultats pourraient ne pas être disponibles avant 4 ans) :

- Ces résultats seront mis dans votre dossier médical.
- Ces résultats génétiques peuvent signaler l'existence d'un risque chez les personnes qui vous sont apparentées, et donc avoir des incidences sur votre famille.
- Vous devrez peut-être subir de nouveaux tests.
- Certains résultats pourraient évoquer des inquiétudes justifiant de recevoir un soutien psychologique.

| <ul> <li>Je souhaite être informérésultats susceptibles de m</li></ul> | e par la médecin-investigatrice/le médecin-investigateur des<br>e concerner : |
|---|---|
| <ul><li>Je souhaite que ma/mon m<br/>concerner :</li><li>Oui</li><li>Non</li></ul> | édecin traitant·e soit informé·e des résultats susceptibles de me |
| <u>Médecin Traitant·e : Nom, Prénom</u> | |
| Si pas de médecin traitant·e : autre | e personne de contact : Nom, Prénom |
| Lieu, date | Signature de la participante / du participant |
| avoir expliqué à la participante/au p<br>satisfaire à toutes les obligations er<br>Si je devais prendre connaissance | tigatrice/du médecin-investigateur: Par la présente, j'atteste participant la nature, l'importance et la portée du projet. Je déclare n' relation avec ce projet conformément au droit suisse en vigueur. e, à quelque moment que ce soit durant la réalisation du projet, ur le consentement de la participante/du participant à prendre part ner immédiatement. |
| Lieu, date | Nom et prénom de la médecine-investigatrice/du médecin-investigateur en caractères d'imprimerie. |
| | Signature de la médecine-investigatrice/du médecin-investigateur |



# @neurIST : informatique biomédicale intégrée pour la gestion des anévrismes cérébraux Ce projet est organisé par : Hôpitaux Universitaire de Genève

Madame, Monsieur,

Nous vous proposons ici de nous accorder votre consentement pour la participation de la patiente/du patient à notre projet.

La présente notice d'information est destinée à être lue en parallèle avec la notice générale d'information destinée aux participant·e·s, qui doit également vous avoir été remise. Cette feuille d'information ne décrit que les points spécifiques aux tests génétiques.

# 1. Objectifs de l'étude génétique

Des résultats préliminaires publiés dans la littérature montrent que des facteurs génétiques, en parallèle des facteurs environnementaux, pourraient contribuer à l'apparition et au développement des anévrismes, cependant leurs rôles précis ne sont pas encore élucidés. Le but des tests génétiques au sein de notre étude @neurIST est donc d'identifier les gènes qui seraient impliqués dans les anévrismes cérébraux.

## 2. Déroulement pour les participants

Une analyse génétique couvrant tout le génome de la patiente/du patient sera effectuée sur l'échantillon sanguin de la patiente/du patient prélevé lors d'une consultation avec le clinicien en charge de la patiente/du patient ou avec la médecin-investigatrice/le médecin-investigateur.

Les gènes des patient·e·s présentant des anévrismes cérébraux seront comparés aux gènes de sujets contrôles (participant·e·s inclus·e·s dans l'étude en tant que « Membre de la famille » ou en tant que « Volontaire·s sain·e·s ») afin de découvrir des variantes dans le génome des patients qui pourraient être associées à une susceptibilité plus importante pour les anévrismes cérébraux.

Si la patiente/le patient fait partie de l'étude familiale, l'ensemble de son génome sera comparé à celui d'autres membres de sa famille afin également de découvrir des gènes candidats liés aux anévrismes.

Ces gènes candidats seront ensuite utilisés pour tester les échantillons de sang remis par des patient·e·s présentant un anévrisme. Les résultats de ces expériences seront placés dans des bases de données informatisées sécurisées. Leur analyse pourrait prendre jusqu'à dix ans.

#### 3. Risques

Les risques associés à cette étude sont ceux liés à la réalisation d'une prise de sang (risque infectieux faible, hématome) et l'utilisation d'un réseau informatique pour le transfert des données dont la sécurité ne peut jamais être totalement garantie.

Nous nous efforcerons de rendre les prises de sang aussi peu douloureuses que possible et mettrons en place des mesures de sécurité pour tous nos transferts de données codées.

Un risque associé à l'étude génétique est la découverte fortuite d'une anomalie associée à une maladie connue. Si certains résultats issus de cette étude génétique étaient susceptibles d'engendrer des inquiétudes chez la patiente/le patient, nous proposerons un soutien psychologique.

## 4. Découvertes pendant l'étude génétique

Toute découverte survenant durant l'étude et pertinente pour la santé de la patiente/du patient vous sera communiquée. Si vous ne souhaitez pas obtenir ce type d'information, veuillez en aviser la médecin-investigatrice/le médecin-investigateur.

Ces résultats génétiques peuvent avoir un impact sur la famille de la patiente/du patient, avec laquelle elle/il partage certains gènes. Si ce cas de figure survient, nous discuterons avec vous sur comment informer les autres membres de la famille.

Version du 12.07.2022



Si la patiente/le patient participe à l'étude familiale, les tests pourraient également révéler des cas de non-paternité; ces résultats ne seront communiqués ni à la patiente/au patient, ni à vous-même ni aux autres membres de la famille de la patiente/du patient.

## 5. Confidentialité des données et des échantillons biologiques

D'une manière générale, le traitement et codages des données, ainsi que la protection des données et des échantillons sont similaires à ce qui est décrit dans la lettre d'information générale qui vous a été donnée dans le cadre du projet @neurIST.

Concernant le cas particulier de la protection des données en cas d'analyses génétiques : Dès lors que l'on procède à un relevé, un enregistrement ou une transmission de données issues des échantillons dans le cadre de la recherche génétique, il existe des risques liés à la confidentialité (p. ex., la possibilité d'identifier la patiente/le patient), en particulier concernant les informations sur son matériel génétique. Ces risques ne peuvent pas être totalement exclus et augmentent avec la quantité de données pouvant être appariées, notamment si la patiente/le patient publie elle/lui-même des données génétiques sur Internet (p. ex. à des fins de recherche généalogique). Les informations relatives à son matériel génétique peuvent également être importantes pour les membres de sa famille ou sa planification familiale. Le promoteur prend toutes les mesures nécessaires pour réduire le plus possible les risques liés à la confidentialité.

## 6. Participation à l'étude génétique et retrait de l'étude

Vous pouvez décider que la patiente/le patient ne participe pas à l'étude génétique @neurIST, tout en fournissant d'autres informations à l'étude. Si vous décidez que la patiente/le patient ne participe pas, cela ne changera rien à sa prise en charge médicale, de son anévrisme le cas échéant. Vous n'avez pas à justifier vos décisions.

Vous pouvez à tout moment retirer la patiente/le patient de l'étude génétique si vous le souhaitez. Vous n'avez pas à justifier vos décisions. Les données médicales recueillies jusque-là seront tout de même analysées car une fois intégrées à la base de données leur destruction devient impossible. Vous pourrez choisir si vous souhaitez que :

- les données soient gardées sous forme codée (codée signifie que le matériel biologique et les données ne peuvent être mis en relation avec la patiente/le patient qu'au moyen d'une clé) ou anonymisée (anonymisée signifie que le code reliant les données à la patiente/au patient sera effacé, plus personne ne pourra savoir que ces données et ces échantillons sont ceux de la patiente/du patient);
- les échantillons biologiques soient conservés ou détruits.

## 7. Interlocuteurs

Vous pouvez à tout moment poser vos questions et demander toutes les précisions nécessaires en vous adressant au :

Dr Philippe Bijlenga, responsable du projet : 079 204 40 43

Secrétariat du Dr Bijlenga : 022 372 34 26 En écrivant à aneurist : ccc@hcuge.ch

En consultant notre site internet : www.aneurist.org



# Déclaration de consentement pour l'étude génétique @neurIST

Veuillez lire attentivement ce formulaire. N'hésitez pas à poser des questions lorsque vous ne comprenez pas quelque chose ou que vous souhaitez avoir des précisions. Votre consentement écrit est nécessaire pour la participation de la patiente/du patient au projet.

| Numéro BASEC du projet :<br>(après soumission à la commission d'éthique<br>compétente) : | 2022-00426 |
|---|---|
| Titre de l'étude :<br>(titre scientifique et titre usuel) | @neurIST : informatique biomédicale intégrée pour la gestion des anévrismes cérébraux |
| Institution responsable : (adresse complète) : | Hôpitaux Universitaire de Genève<br>Rue Micheli-du-Crest 24<br>1211 Genève 14 |
| Lieu de réalisation du projet : | Genève, Suisse |
| Directeur du projet sur le site : (nom et prénom en caractères d'imprimerie) : | Dr Philippe Bijlenga |
| Participant / participante :<br>(nom et prénom en caractères d'imprimerie) :<br>Date de naissance : | |

- En ma qualité de proche ou de représentant e légal e de la patiente/du patient susmentionné e, je déclare avoir été informé e par la médecin-investigatrice/le médecin-investigateur soussigné e, oralement et par écrit, des objectifs et du déroulement du projet ainsi que des effets présumés, des avantages, des inconvénients possibles et des risques éventuels.
- Je confirme prendre la décision dans le sens du proche ou de la personne placée sous ma responsabilité, à savoir, qu'elle/qu'il participe au projet de recherche. En son nom, j'accepte les informations écrites et orales. J'ai eu suffisamment de temps pour prendre ma décision.
- J'ai reçu les réponses aux questions que j'ai posées en relation avec la participation de la patiente/du patient à ce projet. Je conserve la feuille d'information et reçois une copie de ma déclaration de consentement écrite.
- J'accepte que les spécialistes compétent·e·s de la direction de ce projet et de la commission d'éthique compétente puissent consulter les données non codées de la patiente/du patient afin de procéder à des contrôles et des inspections, à condition toutefois que la confidentialité de ces données soit strictement assurée.
- Si la patiente/le patient bénéficie / devais bénéficier d'un traitement médical en dehors de l'institution responsable de ce projet, j'accepte que le médecin responsable du projet contacte la/le médecin traitant·e de la patiente/du patient et que celui-ci lui fournisse des données médicales concernant la patiente/le patient pouvant être pertinentes pour ce projet.
- Je sais que les données personnelles et les échantillons peuvent être transmis à des fins de recherche dans le cadre de ce projet et uniquement sous une forme codée. Le promoteur assure une protection des données conforme aux normes et exigences Suisses.
- Au nom de la patiente/du patient, je peux, à tout moment et sans avoir à me justifier, révoquer son consentement à la participation, sans que cette décision n'ait de répercussions défavorables sur la suite de sa prise en charge. Les données et les échantillons recueillis jusqu'au retrait seront cependant analysés dans le cadre du projet.
- Je suis informé·e que les HUG sont responsables des dommages éventuels imputables au projet.
- Je suis conscient e que les obligations mentionnées dans la feuille d'information destinée aux participant e s doivent être respectées pendant toute la durée du projet. La médecin-



investigatrice/le médecin-investigateur peut exclure la patiente/le patient du projet à tout moment dans l'intérêt de ma santé.

■ Je consens que la patiente/le patient sus-mentionné e participe à cette étude.

Veuillez étudier les points suivants avant de décider si vous souhaitez être informé·e des résultats de la recherche susceptibles d'être pertinents pour la santé de la patiente/du patient (ces résultats pourraient ne pas être disponibles avant 4 ans) :

- Ces résultats seront mis dans le dossier médical de la patiente/du patient.
- Ces résultats peuvent signaler l'existence d'un risque chez les personnes qui sont apparentées à la patiente/au patient, et donc avoir des incidences sur sa famille.
- La patiente/le patient devra peut-être subir de nouveaux tests.
- Certains résultats pourraient évoquer des inquiétudes justifiant de recevoir un soutien psychologique.

| | e par la médecin-investigatrice/le médecin-investigateur des<br>ncerner la patiente/le patient : |
|---|---|
| <ul> <li>Je souhaite que la/le médec<br/>susceptibles de la/le concert<br/>Oui<br/>Non</li> </ul> | in traitant·e de la patiente/du patient soit informé·e des résultats<br>ner : |
| Médecin Traitant·e : Nom, Prénom | |
| Si pas de médecin traitant·e : autre | personne de contact : Nom, Prénom |
| Lieu, date | Relation avec la patiente/le patient : Personne désignée dans les directives anticipées ou dans un mandat pour cause d'inaptitude Curateur/Curatrice Conjoint·e ou son/sa partenaire enregistré·e et fournissant une assistance personnelle régulière Personne faisant ménage commun avec le/la participant·e et fournissant une assistance personnelle régulière Descendant·e et fournissant une assistance personnelle régulière Père/Mère et fournissant une assistance personnelle régulière Frère/Soeur et fournissant une assistance personnelle régulière Frère/Soeur et fournissant une assistance personnelle régulière |



| S | ignature de la/du proche ou de la/du représentant⋅e légal⋅e : |
|---|---------------------------------------------------------------|

Attestation de la médecin-investigatrice/du médecin-investigateur : Par la présente, j'atteste avoir expliqué au proche ou à la/au représentant·e légal·e du/de la participant·e la nature, l'importance et la portée du projet. Je déclare satisfaire à toutes les obligations en relation avec ce projet conformément au droit en vigueur. Si je devais, à quelque moment que ce soit durant la réalisation du projet, prendre connaissance d'éléments susceptibles d'influer sur le consentement de la participante/du participant à prendre part au projet, je m'engage à en informer immédiatement sa/son proche ou sa/son représentant·e légal·e.

| Lieu, date | Nom et prénom de la médecine-investigatrice/du investigateur en caractères d'imprimerie. | médecin- |
|---|---|---|
| | Signature de la médecine-investigatrice/du investigateur | médecin- |



# Déclaration de consentement écrite pour la réutilisation de données et d'échantillons biologiques

| Numéro BASEC du projet de recherche (après soumission à la commission d'éthique compétente) : | 2022-00426 |
|---|---|
| Titre<br>(scientifique et usuel) : | @neurlST : informatique biomédicale intégrée pour la gestion des anévrismes cérébraux |
| Participante / Participant :<br>Nom et prénom en caractères d'imprimerie :<br>Date de naissance : | |

J'accepte que mes données (génétiques) et mon matériel biologique obtenus dans le cadre de ce projet puissent être réutilisés à des fins de recherche médicale. Cela signifie que le matériel biologique sera conservé dans une biobanque et ultérieurement exploité pour une durée indéfinie, tant que je ne retire pas mon consentement, dans le cadre de futurs projets de recherche.

Je sais que mon matériel biologique et que la liste d'identification sont gardés dans un lieu sûr. Les données et le matériel biologique peuvent être envoyés à des fins d'analyse à une autre banque de données/biobanque située en Suisse ou à l'étranger, à condition qu'elle obéisse à des normes et exigences au moins équivalentes aux normes et exigences Suisses. Toutes les dispositions légales relatives à la protection des données sont respectées.

Je donne mon accord de façon volontaire et je peux à tout moment revenir sur ma décision. Si je reviens sur ma décision, mes données seront gardées sous forme codée (codée signifie que mon matériel biologique et mes données ne peuvent être mis en relation avec ma personne qu'au moyen d'une clé) ou anonymisée (anonymisée signifie que le code reliant mes données à ma personne sera effacé, plus personne ne pourra savoir que ces données et ces échantillons sont les miens). Je déciderai aussi si mon matériel biologique doit être détruit ou conservé. Je dois simplement en informer la médecin-investigatrice/le médecin-investigateur. Je n'ai pas à justifier ma décision.

Je sais que si je choisi que mes données soient rendues anonymes, je ne pourrai plus être informé e des éventuelles découvertes fortuites.

Généralement, les données et le matériel biologique sont exploités de manière globale et les résultats sont publiés de manière synthétique. Il se peut que je sois contacté·e si l'analyse des données révèle une découverte pertinente pour ma santé. Si je ne souhaite pas en être informé·e, il m'incombe d'en aviser la médecin-investigatrice/le médecin-investigateur.

Je renonce à tout droit d'exploitation commerciale sur le matériel biologique qui m'a été prélevé et sur mes données.

| 0 | J'accepte que mes données et mes échantillons biologiques puissent être réutilisés à des fins de recherche médicale. Oui Non |
|---|---|
| 0 | Si oui, je souhaite que mes données et mes échantillons soient réutilisés sous forme : Codée Anonymisée |




| <ul> <li>Je souhaite être informéries de m</li> <li>Oui</li> <li>Non</li> </ul> | e par la médecin-investigatrice/le médecin-investigateur des le concerner : |
|---|---|
| <ul><li>Je souhaite que ma/mon m<br/>concerner :</li><li>Oui</li><li>Non</li></ul> | nédecin traitant·e soit informé·e des résultats susceptibles de me |
| <u>Médecin Traitant·e : Nom, Prénom</u> | <u>l</u> |
| Si pas de médecin traitant·e : autre | e personne de contact : Nom, Prénom |
| Lieu, date | Signature de la participante / du participant |
| avoir expliqué à la participante/au p<br>satisfaire à toutes les obligations en<br>Si je devais prendre connaissance | ctigatrice/du médecin-investigateur: Par la présente, j'atteste participant la nature, l'importance et la portée du projet. Je déclare n relation avec ce projet conformément au droit suisse en vigueur. e, à quelque moment que ce soit durant la réalisation du projet, ur le consentement de la participante/du participant à prendre part ner immédiatement. |
| Lieu, date | Nom et prénom de la médecine-investigatrice/du médecin-investigateur en caractères d'imprimerie. |
| | Signature de la médecine-investigatrice/du médecin-<br>investigateur |




# Déclaration de consentement écrite pour la réutilisation de données et d'échantillons biologiques

| Numéro BASEC du projet de recherche (après soumission à la commission d'éthique compétente) : | 2022-00426 |
|---|---|
| Titre<br>(scientifique et usuel) : | @neurlST : informatique biomédicale intégrée pour la gestion des anévrismes cérébraux |
| Participante / Participant :<br>Nom et prénom en caractères d'imprimerie :<br>Date de naissance : | |

J'accepte que les données (génétiques) et le matériel biologique de la patiente/du patient obtenus dans le cadre de ce projet puissent être réutilisés à des fins de recherche médicale. Cela signifie que le matériel biologique sera conservé dans une biobanque et ultérieurement exploité pour une durée indéfinie, tant que la patiente/le patient ou même ne retire pas le consentement, dans le cadre de futurs projets de recherche.

Je sais que le matériel biologique et que la liste d'identification sont gardés dans un lieu sûr. Les données et le matériel biologique peuvent être envoyés à des fins d'analyse à une autre banque de données/biobanque située en Suisse ou à l'étranger, à condition qu'elle obéisse à des normes et exigences au moins équivalentes aux normes et exigences Suisses. Toutes les dispositions légales relatives à la protection des données sont respectées.

Je donne mon accord de façon volontaire et je peux à tout moment revenir sur ma décision. Si je reviens sur ma décision, les données de la patiente/du patient seront gardées sous forme codée (codée signifie que le matériel biologique et les données de la patiente/du patient ne peuvent être mis en relation avec sa personne qu'au moyen d'une clé) ou anonymisée (anonymisée signifie que le code reliant les données à la patiente/au patient sera effacé, plus personne ne pourra savoir que ces données et ces échantillons sont les siens). Je déciderai aussi si le matériel biologique de la patiente/du patient doit être détruit ou conservé. Je dois simplement en informer la médecininvestigatrice/le médecin-investigateur. Je n'ai pas à justifier ma décision.

Je sais que si je choisi que les données de la patiente/du patient soient rendues anonymes, je ne pourrai plus être informé·e des éventuelles découvertes fortuites.

Généralement, les données et le matériel biologique sont exploités de manière globale et les résultats sont publiés de manière synthétique. Il se peut que je sois contacté·e si l'analyse des données révèle une découverte pertinente pour la santé de la patiente/du patient. Si je ne souhaite pas en être informé·e, il m'incombe d'en aviser la médecin-investigatrice/le médecin-investigateur.

Je renonce à tout droit d'exploitation commerciale sur le matériel biologique qui a été prélevé et sur les données de la patiente/du patient.

| 0 | J'accepte que les données et les échantillons biologiques de la patiente/du patient puissent |
|---|---|
| | être réutilisés à des fins de recherche médicale. |
| | Oui |
| | Non |

 Si oui, je souhaite que les données et les échantillons de la patiente/du patient soient réutilisés sous forme :


| Hôpitaux<br>Universitaires<br>Genève | |
|---|---|
| Codée Anony | |
| résultats susceptibles de co<br>Oui<br>Non | e par la médecin-investigatrice/le médecin-investigateur des<br>ncerner la patiente/le patient:<br>n traitant·e de la patiente/du patient soit informé·e des résultats<br>ner : |
| <br>Médecin Traitant·e : Nom, Prénom | |
| Si pas de médecin traitant·e : autre | personne de contact : Nom, Prénom |
| Lieu, date | Nom et prénom en caractères d'imprimerie |
| | Relation avec la patiente/le patient : Personne désignée dans les directives anticipées ou dans un mandat pour cause d'inaptitude Curateur/Curatrice Conjoint·e ou son/sa partenaire enregistré·e et fournissant une assistance personnelle régulière Personne faisant ménage commun avec le/la participant·e et fournissant une assistance personnelle régulière Descendant·e et fournissant une assistance personnelle régulière Père/Mère et fournissant une assistance personnelle régulière Frère/Soeur et fournissant une assistance personnelle régulière Signature de la/du proche ou de la/du représentant·e légal·e : |

Attestation de la médecin-investigatrice/du médecin-investigateur : Par la présente, j'atteste avoir expliqué au proche ou à la/au représentant·e légal·e du/de la participant·e la nature, l'importance et la portée du projet. Je déclare satisfaire à toutes les obligations en relation avec ce




projet conformément au droit en vigueur. Si je devais, à quelque moment que ce soit durant la réalisation du projet, prendre connaissance d'éléments susceptibles d'influer sur le consentement de la participante/du participant à prendre part au projet, je m'engage à en informer immédiatement sa/son proche ou sa/son représentant·e légal·e.

| Lieu, date | Nom et prénom de la médecine-investigatrice/du médecin-<br>investigateur en caractères d'imprimerie. |
|---|---|
| | Signature de la médecine-investigatrice/du médecin-<br>investigateur : |




# Déclaration de retrait de consentement de l'étude @neurIST : informatique biomédicale intégrée pour la gestion des anévrismes cérébraux

Veuillez lire attentivement ce formulaire. N'hésitez pas à poser des questions lorsque vous ne comprenez pas quelque chose ou que vous souhaitez avoir des précisions.

| Numéro BASEC du projet de recherche<br>(après soumission à la commission<br>d'éthique compétente) : | 2022-00426 |
|---|---|
| Titre (scientifique et usuel) : | @neurIST : informatique biomédicale intégrée pour la gestion des anévrismes cérébraux |
| Institution responsable<br>(responsable du projet et adresse<br>complète) : | Hôpitaux Universitaire de Genève<br>Rue Micheli-du-Crest 24<br>1211 Genève 14 |
| Lieu de réalisation : | Genève, Suisse |
| Responsable du projet sur le site :<br>Nom et prénom en caractères d'imprimerie : | Dr Philippe Bijlenga |
| Participante / Participant :<br>Nom et prénom en caractères d'imprimerie :<br>Date de naissance : | |
| mes consentement s pour ma participation Retrait du conser | de recherche sus-mentionné du retrait de mon / de<br>à ce projet.<br>Itement général au projet @neurIST<br>Itement pour l'étude génétique @neurIST |
| | issues de l'analyse de mon matériel biologique<br>inservées car une fois intégrées à la base de données |
| J'accepte que mes échantillons biologiquéchantillons seront alors détruits) : Oui Non | ues soient conservés (dans le cas contraire, vos |
| en relation avec r<br>Anonymisée (le c<br>plus personne ne<br>sont les miens). | ériel biologique et mes données ne pouront être mis<br>na personne qu'au moyen d'une clé).<br>ode reliant mes données à ma personne sera effacé,<br>e pourra savoir que ces données et ces échantillons<br>Je sais que si je choisi que mes données soient<br>es, je ne pourrai plus être informé e des éventuelles |

Version du 12.07.2022



| Je souhaite que lien e | ntre mes données cliniques et génétiques soit supprimé :<br>Oui<br>Non |
|---|---|
| Lieu, date | Signature de la participante/du participant |
| Attestation de la médecin-investigatrice / du médecin-investigateur : Lieu, date Nom et prénom de la médecine-investigatrice/du minvestigateur en caractères d'imprimerie. | |
| | Signature de la médecine-investigatrice/du médecin-investigateur |





# Déclaration de retrait de consentement de l'étude @neurIST : informatique biomédicale intégrée pour la gestion des anévrismes cérébraux

Veuillez lire attentivement ce formulaire. N'hésitez pas à poser des questions lorsque vous ne comprenez pas quelque chose ou que vous souhaitez avoir des précisions.

| Numéro BASEC du projet de recherche<br>(après soumission à la commission<br>d'éthique compétente) : | 2022-00426 |
|---|---|
| Titre<br>(scientifique et usuel) : | @neurIST : informatique biomédicale intégrée pour la gestion des anévrismes cérébraux |
| Institution responsable<br>(responsable du projet et adresse<br>complète) : | Hôpitaux Universitaire de Genève<br>Rue Micheli-du-Crest 24<br>1211 Genève 14 |
| Lieu de réalisation : | Genève, Suisse |
| Responsable du projet sur le site :<br>Nom et prénom en caractères d'imprimerie : | Dr Philippe Bijlenga |
| Participante / Participant :<br>Nom et prénom en caractères d'imprimerie :<br>Date de naissance : | |
| consentement s de la patiente/du patient s Retrait du conser Retrait du conser Les données médicales et les valeurs | ojet de recherche sus-mentionné du retrait du/des<br>us-mentionné e pour sa participation à ce projet.<br>ntement général au projet @neurIST<br>ntement pour l'étude génétique @neurIST<br>issues de l'analyse de son matériel biologique |
| (échantillons de sang, tissus, etc.) seront co<br>leur destruction devient impossible. | onservées car une fois intégrées à la base de données |
| J'accepte que les échantillons biologique conservés (dans le cas contraire, les échar Oui Non | s de la patiente/du patient sus-mentionné·e soient<br>ntillons seront alors détruits) : |
| gardés sous forme : Codée (le matéric relation avec la partic Anonymisée (le compersonne sera é données et ces ée ses données so | lons de la patiente/du patient sus-mentionné·e soient el biologique et les données ne pouront être mis en atiente/le patient qu'au moyen d'une clé). ode reliant les données de la patiente/du patient à sa effacé, plus personne ne pourra savoir que ces chantillons sont les siens). Je sais que si je choisi que ient rendues anonymes, je ne pourrai plus être entuelles découvertes fortuites. |

Version du 12.07.2022



| Je souhaite que lien entre les c<br>Oui<br>Non | données cliniques et génétiques soit supprimé : |
|---|---|
| Lieu, date | Nom et prénom en caractères d'imprimerie |
| | Relation avec la patiente/le patient : |
| | Personne désignée dans les directives anticipées ou dans un mandat pour cause d'inaptitude |
| | Curateur/Curatrice Conjoint·e ou son/sa partenaire enregistré·e et fournissant une assistance personnelle régulière |
| | <ul> <li>☐ Personne faisant ménage commun avec le/la participant·e et fournissant une assistance personnelle régulière</li> <li>☐ Descendant·e et fournissant une assistance personnelle régulière</li> </ul> |
| | Père/Mère et fournissant une assistance personnelle régulière |
| | Frère/Soeur et fournissant une assistance personnelle régulière |
| | Signature de la/du proche ou de la/du représentant·e légal·e : |
| avoir expliqué au proche ou à<br>l'importance et la portée du projet.<br>projet conformément au droit en<br>réalisation du projet, prendre conr | tigatrice/du médecin-investigateur : Par la présente, j'atteste la/au représentant·e légal·e du/de la participant·e la nature, Je déclare satisfaire à toutes les obligations en relation avec ce vigueur. Si je devais, à quelque moment que ce soit durant la naissance d'éléments susceptibles d'influer sur le consentement prendre part au projet, je m'engage à en informer immédiatement tant·e légal·e. |
| Lieu, date | Nom et prénom de la médecine-investigatrice/du médecin-<br>investigateur en caractères d'imprimerie. |
| | Signature de la médecine-investigatrice/du médecin-investigateur |